CLINICAL TRIAL: NCT02522299
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Efficacy and Changes in Induced Sputum and Blood Biomarkers Following Daily Repeat Doses of Inhaled GSK2269557 for 12 Weeks in Adult Subjects Diagnosed With an Acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Evaluate the Safety, Efficacy and Changes in Induced Sputum and Blood Biomarkers Following Daily Repeat Doses of Inhaled GSK2269557 in Chronic Obstructive Pulmonary Disease (COPD) Subjects With Acute Exacerbation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201928; 2015-003696-30 (EudraCT Number)
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: double-blind; PI3Kdelta; GSK2269557; exacerbation; Chronic Obstructive Pulmonary Disease; randomised; placebo-controlled
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nemiralisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK2269557 1000 microgram (mcg) (Experimental): Subjects will receive 2 inhalations of GSK2269557 (30 seconds apart, 2 x 500 mcg, total dose of 1000 mcg) once daily for 84 consecutive days via DISKUS™ device.
  Interventions: Drug: GSK2269557; Device: DISKUS
- Placebo via DISKUS (Placebo Comparator): Subjects will receive 2 inhalations of placebo once daily for 84 days via DISKUS device.
  Interventions: Drug: Placebo; Device: DISKUS
- GSK2269557 700 mcg (Experimental): Subjects will receive 2 inhalations of GSK2269557 700 mcg once daily for 84 consecutive days via ELLIPTA.
  Interventions: Device: ELLIPTA
- Placebo via ELLIPTA (Placebo Comparator): Subjects will receive Placebo once daily for 84 consecutive days via ELLIPTA.
  Interventions: Drug: Placebo; Device: ELLIPTA

INTERVENTIONS:
Drug: GSK2269557 — GSK2269557 500 mcg blended with lactose per blister and will be administered using a DISKUS dry powder inhaler device. Since GSK2269557 will no longer be manufactured for use with the DISKUS device, it will be replaced with ELLIPTA Device. Subjects will receive GSK2269557 700 mcg once daily for 84 consecutive days via ELLIPTA.
  Arms: GSK2269557 1000 microgram (mcg)
Drug: Placebo — Lactose will be administered using a DISKUS and ELLIPTA dry powder inhaler device
  Arms: Placebo via DISKUS; Placebo via ELLIPTA
Device: DISKUS — It is multi-dose dry powder inhaler containing one foil strip of drug with 60 blisters
  Arms: GSK2269557 1000 microgram (mcg); Placebo via DISKUS
Device: ELLIPTA — It is multi-dose dry powder inhaler containing one foil strip of drug with 30 blisters
  Arms: GSK2269557 700 mcg; Placebo via ELLIPTA

SUMMARY:
The purpose of this study is to evaluate specific alterations in immune cell mechanisms related to neutrophil function as detected by PI3Kdelta-dependent changes in messenger ribonucleic acid (mRNA) extracted from induced sputum in patients experiencing an exacerbation of COPD, with or without treatment with GSK2269557. The efficacy of treatment with GSK2269557 will also be measured using functional respiratory imaging (FRI) and spirometry. This is a randomised, double-blind, placebo-controlled, parallel-group study. The study consisted of Screening Phase (up to 3 days prior to Day 1), Treatment Phase (Days 1 to 84) and Follow phase (7 to 14 days after last dose). The total duration of the study is 13-14 weeks including the screening visit. DISKUS TM and ELLIPTA TM are registered trademark of GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years of age inclusive, at the time of signing the informed consent.
* The subject has a confirmed and established diagnosis of COPD, as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines for at least 6 months prior to entry.
* The subject is able to produce >100 milligram (mg) of sputum at screening for processing, (ie, total weight of sputum plugs).
* The subject has a post-bronchodilator FEV1/FVC <0.7 and FEV1 <=80 % of predicted.
* Disease severity: Acute exacerbation of COPD requiring an escalation in therapy to include both corticosteroid and antibiotics. Acute exacerbation to be confirmed by an experienced physician and represent a recent change in at least two major and one minor symptoms, one major and two minor symptoms, or all 3 major symptoms. Major symptoms: Subjective increase in dyspnea; Increase in sputum volume; Change in sputum colour. Minor symptoms: Cough; Wheeze; Sore throat
* The subject is a smoker or an ex-smoker with a smoking history of at least 10 pack years (pack years = [cigarettes per day smoked/20 x number of years smoked]).
* Body weight >= 45 kilogram (kg) and body mass index (BMI) within the range 16 to 35 kilogram per meter square (kg/m^2) (inclusive)
* Male
* Female subject: is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: (1)Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea. Females whose menopausal status is in doubt will be required to use, or have been using, one of the highly effective contraception methods as specified below from 30 days prior to the first dose of study medication and until completion of the follow-up visit. 2)Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until completion of the follow-up visit. GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP. This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis. 1) Contraceptive subdermal implant that meets GSK standard criteria including a <1% rate of failure per year, as stated in the product label. 2) Intrauterine device or intrauterine system that meets GSK standard criteria including a <1% rate of failure per year, as stated in the product label. 3) Oral Contraceptive, either combined or progestogen alone. 4) Injectable progestogen. 5) Contraceptive vaginal ring. 6) Percutaneous contraceptive patches. 7) Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. 8) Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository). These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. Specific inclusion criteria for Male subjects with female partners of reproductive potential is outlined below: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until after the completion of the follow up visit. 1) Vasectomy with documentation of azoospermia. 2) Male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant that meets GSK standard criteria including a <1% rate of failure per year, as stated in the product label. Intrauterine device or intrauterine system that meets GSK standard criteria including a <1% rate of failure per year, as stated in the product label. Oral Contraceptive, either combined or progestogen alone. Injectable progestogen. Contraceptive vaginal ring. Percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* To avoid recruitment of subjects with a severe COPD exacerbation, the presence of any one of the following severity criteria will render the subject ineligible for inclusion in the study: Need for invasive mechanical ventilation (short term [<48 hour] Non-invasive ventilation [NIV] or continuous positive airway pressure [CPAP] is acceptable); Haemodynamic instability or clinically significant heart failure; Confusion; Clinically significant pneumonia, identified by chest X-ray at screening, and as judged by the Investigator.
* Subjects who have current medical conditions or diseases that are not well controlled and, which as judged by the Investigator, may affect subject safety or influence the outcome of the study. (Note: Patients with adequately treated and well controlled concurrent medical conditions (e.g. hypertension or noninsulin-dependent diabetes mellitus [NIDDM]) are permitted to be entered into the study).
* Subject has a diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, pulmonary fibrosis, asthma or any other respiratory condition that might, in the opinion of the investigator, compromise the safety of the subject or affect the interpretation of the results.
* ALT >2xupper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the exclusion criteria, outside of the reference range for the population being studied may be included if the Investigator [in consultation with the GSK Medical Monitor if required] documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* ECG indicative of an acute cardiac event (e.g. Myocardial Infarction) or demonstrating a clinically significant arrhythmia requiring treatment.
* QTcF > 450 msec or QTcF > 480 msec in subjects with Bundle Branch Block, based on single QTcF value.
* Subjects who have undergone lung volume reduction surgery.
* Subject is currently on chronic treatment with macrolides or long term antibiotics.
* Subject is being treated with long term oxygen therapy (LTOT) (>15 hours/day).
* The subject has been on chronic treatment with anti-Tumour Necrosis Factor (anti-TNF), or any other immunosuppressive therapy (except corticosteroid) within 60 days prior to dosing
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >28 units for males or >21 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof (such as lactose) or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* A known (historical) positive test for human immunodeficiency virus (HIV) antibody.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. NOTE: Because of the short window for screening, treatment with GSK2269557 may start before receiving the result of the hepatitis tests. If subsequently the test is found to be positive, the subject may be withdrawn, as judged by the Principal Investigator in consultation with the Medical Monitor.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Montreal, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20861

REFERENCES:
- [Background] Begg M, Hamblin JN, Jarvis E, Bradley G, Mark S, Michalovich D, Lennon M, Wajdner HE, Amour A, Wilson R, Saunders K, Tanaka R, Arai S, Tang T, Van Holsbeke C, De Backer J, Vos W, Titlestad IL, FitzGerald JM, Killian K, Bourbeau J, Poirier C, Maltais F, Cahn A, Hessel EM. Exploring PI3Kdelta Molecular Pathways in Stable COPD and Following an Acute Exacerbation, Two Randomized Controlled Trials. Int J Chron Obstruct Pulmon Dis. 2021 Jun 3;16:1621-1636. doi: 10.2147/COPD.S309303. eCollection 2021. PMID 34113094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 44 participants with Chronic obstructive pulmonary disease (COPD) were enrolled in this study. The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA.but the 2 treatment arms remained the same i.e. Placebo and GSK2269557 (Nemiralisib [NEMI]).There was no intent to compare two devices.
Pre-assignment Details: As the switch to the ELLIPTA device was intended to be a comparable treatment, the treatment groups Placebo DISKUS and Placebo ELLIPTA were combined as All Placebo treatment group. Similarly, the treatment groups NEMI DISKUS and NEMI ELLIPTA were combined as All NEMI treatment group.
Groups:
- All Placebo: Participants were administered with placebo matching NEMI once daily in the morning before breakfast for 84 consecutive days using DISKUS or ELLIPTA dry powder inhaler (DPI).
- All NEMI: Participants were administered with either NEMI 1000 micrograms (mcg) once daily in the morning using DISKUS DPI or 700 mcg once daily in the morning using ELLIPTA DPI before breakfast for 84 consecutive days
Period: Overall Study
Arm/Group | All Placebo | All NEMI
Started | 22 | 22
Completed | 18 | 21
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI. There was no intent to compare two devices.
Groups:
- Total: Total of all reporting groups
Arm/Group | All Placebo | All NEMI | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (8.20) | 66.1 (7.32) | 65.1 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European Heritage | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Messenger Ribonucleic Acid (mRNA) Transcriptome in Induced Sputum After 12, 28 and 84 Days of Treatment (Selected Probe Sets With Fold Change >1.5 or <-1.5 and p<0.05) in NEMI Treatment Group
Description: Saline-induced sputum samples were collected at the indicated time-points to determine the alterations in previously identified immune cell mechanisms specifically related to neutrophil function by identifying the changes in mRNA transcriptome in induced sputum. Baseline was defined as screening visit. The log2 transformed mRNA intensities for each probe set were analyzed in a separate repeated measures model. Back transformed baseline-adjusted ratios and two-sided unadjusted p-values were calculated for each visit as the specified time-point value/baseline value. These ratios were converted to fold change values; if ratio >= 1 then fold change=ratio or if ratio < 1 then fold change = -1/ratio. Data for pre-specified probe sets that meet the criteria fold change >1.5 or <-1.5 and p<0.05 for All NEMI, All Placebo and All NEMI/All Placebo group is presented in outcome measure 1, 2 and 3 respectively. In the categories column we have included time-point, Probe ID and Gene label.
Time Frame: Baseline (Screening) and Days 12, 28 and 84
Population: All Subjects Population comprised of all randomized participants who received at least one dose of the study treatment.
Measure: Number; unit: Fold change
Arm/Group | All NEMI
Number analyzed (Participants) | 22
Fold change
  Day 12,222834_s_at, GNG12 | 1.78
  Day 12,210390_s_at, CCL15 | 1.72
  Day 12,212294_at, GNG12 | 1.67
  Day 12,226497_s_at, FLT1 | 1.57
  Day 12, 204356_at, LIMK1 | 1.54
  Day 12, 203923_s_at, CYBB | 1.51
  Day 12, 219748_at, TREML2 | -1.51
  Day 12, 1555086_at, STAT5B | -1.51
  Day 12, 211883_x_at, CEACAM1 | -1.51
  Day 12, 224909_s_at, PREX1 | -1.51
  Day 12, 239170_at, ACTR3 | -1.51
  Day 12, 212550_at, STAT5B | -1.52
  Day 12, 202178_at, PRKCZ | -1.52
  Day 12, 219633_at, TTPAL | -1.53
  Day 12, 204285_s_at, PMAIP1 | -1.56
  Day 12, 1555088_x_at, STAT5B | -1.56
  Day 12, 227817_at, PRKCB | -1.57
  Day 12, 205632_s_at, PIP5K1B | -1.58
  Day 12, 202018_s_at, LTF | -1.59
  Day 12, 232763_at, TLN1 | -1.59
  Day 12, 202948_at, IL1R1 | -1.60
  Day 12, 1569830_at, PTPRC | -1.63
  Day 12, 215561_s_at, IL1R1 | -1.69
  Day 12, 228031_at, TTPAL | -1.71
  Day 12, 209498_at, CEACAM1 | -1.75
  Day 12, 204563_at, SELL | -1.87
  Day 12, 205118_at, FPR1 | -1.93
  Day 12, 236172_at, LTB4R | -1.96
  Day 12, 212372_at, MYH10 | -2.12
  Day 28, 244313_at, CR1 | 1.99
  Day 28, 213093_at, PRKCA | 1.53
  Day 28, 205778_at, KLK7 | -1.54
  Day 84, 233694_at, HSPA1L | 1.88
  Day 84, 208304_at, CCR3 | 1.83
  Day 84, 215101_s_at, CXCL5 | 1.82
  Day 84,214974_x_at ,CXCL5 | 1.80
  Day 84, 207852_at, CXCL5 | 1.63
  Day 84, 1555759_a_at, CCL5 | -1.51
  Day 84, 207535_s_at, NFKB2 | -1.53
  Day 84, 234212_at, ACTR2 | -1.57
  Day 84, 207794_at, CCR2 | -1.58
  Day 84, 206978_at, CCR2 | -1.64
  Day 84, 211889_x_at, CEACAM1 | -1.69
  Day 84, 206219_s_at, VAV1 | -1.71
  Day 84, 209498_at, CEACAM1 | -1.72
  Day 84, 206576_s_at, CEACAM1 | -1.75
  Day 84, 211883_x_at, CEACAM1 | -1.76

2. Primary Outcome: Change in mRNA Transcriptome in Induced Sputum After 12, 28 and 84 Days of Treatment (Selected Probe Sets With Fold Change >1.5 or <-1.5 and p<0.05) in Placebo Treatment Group
Description: Saline-induced sputum samples were collected at the indicated time-points to determine the alterations in previously identified immune cell mechanisms specifically related to neutrophil function by identifying the changes in mRNA transcriptome in induced sputum. Baseline was defined as screening visit. The log2 transformed mRNA intensities for each probe set were analysed in a separate repeated measures model. Back transformed baseline-adjusted ratios and two-sided unadjusted p-values were calculated for each visit as the specified time-point value/baseline value. These ratios were converted to fold change values; if ratio >= 1 then fold change=ratio or if ratio < 1 then fold change = -1/ratio. Data for pre-specified probe sets that meet the criteria fold change >1.5 or <-1.5 and p<0.05 for All NEMI, All Placebo and All NEMI/All Placebo group is presented in outcome measure 1, 2 and 3 respectively. In the categories column we have included time-point, Probe ID and Gene label.
Time Frame: Baseline (Screening) and Days 12, 28 and 84
Population: All Subjects Population.
Measure: Number; unit: Fold Change
Arm/Group | All Placebo
Number analyzed (Participants) | 22
Fold Change
  Day 12, 222834_s_at, GNG12 | 2.29
  Day 12, 207852_at, CXCL5 | 1.81
  Day 12, 212294_at, GNG12 | 1.79
  Day 12, 209576_at, GNAI1 | 1.61
  Day 12, 213281_at, JUN | 1.51
  Day 12, 222880_at, AKT3 | 1.51
  Day 12, 205026_at, STAT5B | -1.50
  Day 12, 201783_s_at, RELA | -1.50
  Day 12, 227404_s_at, EGR1 | -1.51
  Day 12, 1552552_s_at,CLEC4C | -1.54
  Day 12, 211823_s_at,PXN | -1.55
  Day 12,206978_at,CCR2 | -1.55
  Day 12,206219_s_at,VAV1 | -1.56
  Day 12,219748_at,TREML2 | -1.56
  Day 12,207794_at,CCR2 | -1.58
  Day 12,211561_x_at,MAPK14 | -1.59
  Day 12,226507_at,PAK1 | -1.59
  Day 12,232068_s_at,TLR4 | -1.60
  Day 12,209282_at,PRKD2 | -1.60
  Day 12,226080_at,SSH2 | -1.61
  Day 12,212550_at,STAT5B | -1.64
  Day 12,212372_at,MYH10 | -1.64
  Day 12,214022_s_at,IFITM1 | -1.66
  Day 12,217484_at,CR1 | -1.67
  Day 12,206244_at,CR1 | -1.68
  Day 12,1552480_s_at,PTPRC | -1.68
  Day 12,1554114_s_at,SSH2 | -1.69
  Day 12,201601_x_at,IFITM1 | -1.75
  Day 12,205842_s_at,JAK2 | -1.75
  Day 12,228603_at, ACTR3 | -1.75
  Day 12,230100_x_at,PAK1 | -1.77
  Day 12,239307_at,MYH11 | -1.88
  Day 12,223750_s_at,TLR10 | -1.88
  Day 12,208488_s_at,CR1 | -1.92
  Day 12,204563_at,SELL | -2.70
  Day 28, 222834_s_at,GNG12 | 1.91
  Day 84,226498_at,FLT1 | 4.10
  Day 84,216598_s_at,CCL2 | 1.75
  Day 84,1562439_at,NCOA3 | 1.52
  Day 84,201087_at,PXN | -1.52
  Day 84,224909_s_at,PREX1 | -1.52
  Day 84,211823_s_at,PXN | -1.53
  Day 84,209615_s_at,PAK1 | -1.54
  Day 84,211561_x_at,MAPK14 | -1.59
  Day 84,203749_s_at,RARA | -1.60
  Day 84,219748_at,TREML2 | -1.61
  Day 84,207008_at,CXCR2 | -1.66
  Day 84,244313_at,CR1 | -1.67
  Day 84,202530_at,MAPK14 | -1.69
  Day 84,228648_at,LRG1 | -1.71
  Day 84,208488_s_at,CR1 | -1.71
  Day 84,228795_at,PRKCB | -1.73
  Day 84,1552480_s_at,PTPRC | -1.76
  Day 84,232068_s_at,TLR4 | -1.77
  Day 84,221060_s_at,TLR4 | -1.78
  Day 84,201601_x_at,IFITM1 | -1.79
  Day 84,202018_s_at,LTF | -1.82
  Day 84,217209_at,CEACAM3 | -1.85
  Day 84,214022_s_at,IFITM1 | -1.89
  Day 84,217552_x_at,CR1 | -1.89
  Day 84,203591_s_at,CSF3R | -1.91
  Day 84,205118_at,FPR1 | -1.92
  Day 84,1553297_a_at,CSF3R | -1.96
  Day 84,204563_at,SELL | -2.23
  Day 84,219669_at,CD177 | -2.47

3. Primary Outcome: Change in Messenger Ribonucleic Acid (mRNA) Transcriptome in Induced Sputum After 12, 28 and 84 Days of Treatment (Selected Probe Sets With Fold Change >1.5 or <-1.5 and p<0.05) in All NEMI/All Placebo Comparison Treatment Group
Description: Saline-induced sputum samples were collected at the indicated time-points to determine the alterations in previously identified immune cell mechanisms specifically related to neutrophil function by identifying the changes in mRNA transcriptome in induced sputum. For each probe set, the log2 transformed mRNA intensities were analyzed in separate repeated measures models. The models included a Treatment, Visit and Treatment*Visit term. The Visit consisted of 4 levels: Screening (Baseline), Day 12, Day 28 and Day 84, and the Treatment consisted of three levels: Null (when Visit = Screening), All Placebo and All NEMI. The fold changes were derived from the back transformed ratio from Baselines as fold change = ratio if ratio is >=1, else if ratio <1 then fold change = -1/ratio. Data for pre-specified probe sets that meet the criteria fold change >1.5 and p<0.05 for All NEMI, All Placebo and All NEMI/All Placebo group is presented in outcome measure 1, 2 and 3 respectively.
Time Frame: Baseline (Screening) and Days 12, 28 and 84
Population: All Subjects Population.
Measure: Number; unit: Fold Change
Groups:
- All NEMI/All Placebo: This arm is a comparison of All NEMI and All Placebo Arm
Arm/Group | All NEMI/All Placebo
Number analyzed (Participants) | 44
Fold Change
  Day 12,200671_s_at,SPTBN1 | -1.74
  Day 12,226342_at,SPTBN1 | -1.89
  Day 12,200672_x_at,SPTBN1 | -1.60
  Day 12,209576_at,GNAI1 | -1.62
  Day 12,202178_at,PRKCZ | -1.55
  Day 28,244313_at,CR1 | 2.75
  Day 28,223750_s_at,TLR10 | 2.66
  Day 28,217552_x_at,CR1 | 2.25
  Day 28,206244_at,CR1 | 2.01
  Day 28,208488_s_at,CR1 | 1.95
  Day 28,232068_s_at,TLR4 | 1.71
  Day 28,1553297_a_at,CSF3R | 1.71
  Day 28,1552798_a_at,TLR4 | 1.68
  Day 28,223943_s_at,GNG2 | 1.63
  Day 28,221060_s_at,TLR4 | 1.58
  Day 28,239695_at,JAK1 | 1.52
  Day 28,234290_x_at,MYH14 | -1.52
  Day 28,1568377_x_at,DEFB124 | -1.52
  Day 28,1555765_a_at,GNG4 | -1.53
  Day 28,201464_x_at,JUN | -1.57
  Day 28,201465_s_at,JUN | -1.68
  Day 28,239381_at,KLK7 | -1.69
  Day 28,205778_at,KLK7 | -1.71
  Day 28,213281_at,JUN | -1.72
  Day 84,208304_at,CCR3 | 2.52
  Day 84,1553297_a_at,CSF3R | 2.25
  Day 84,203591_s_at,CSF3R | 1.98
  Day 84,221060_s_at,TLR4 | 1.83
  Day 84,202530_at,MAPK14 | 1.77
  Day 84,244313_at,CR1 | 1.60
  Day 84,203872_at,ACTA1 | 1.53
  Day 84,216944_s_at,ITPR1 | -1.51
  Day 84,215195_at,PRKCA | -1.66
  Day 84,226498_at,FLT1 | -5.18

4. Secondary Outcome: Change From Baseline in Specific Imaging Airway Volume (siVaw) at Functional Residual Capacity (FRC) and Total Lung Capacity (TLC) for Individual Lobes
Description: siVaw was measured at FRC and TLC. Data was collected at longitudinal time points (Untrimmed data): Baseline (Screening), Day 12 & Day 28 and at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For Untrimmed data and SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (n=X1, X2 in the category title). This table presents the untrimmed data (in rows with categories containing untrimmed), SCRD12 scan trim pair data (in rows with categories containing Scan Trimmed and Day 12) and SCRD28 scan trim pair data (in rows with categories containing Scan Trimmed and Day 28) only.
Time Frame: Baseline (Screening), Days 12 and 28
Population: All Subjects Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters per Liter
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters per Liter
  FRC,Scan Trimmed,Right Upper,Day 12,n=17,16: number analyzed (Participants) | 17 | 16
  FRC,Scan Trimmed,Right Upper,Day 12,n=17,16 | 1.020 [0.854 to 1.217] | 1.038 [0.880 to 1.225]
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18 | 1.027 [0.838 to 1.258] | 1.030 [0.924 to 1.147]
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17 | 0.970 [0.798 to 1.180] | 0.993 [0.857 to 1.151]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19 | 1.008 [0.779 to 1.304] | 1.053 [0.937 to 1.184]
  FRC,Scan Trimmed,Right Middle,Day 12,n=17,16: number analyzed (Participants) | 17 | 16
  FRC,Scan Trimmed,Right Middle,Day 12,n=17,16 | 1.294 [0.904 to 1.852] | 1.008 [0.856 to 1.188]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18 | 1.071 [0.773 to 1.484] | 0.973 [0.865 to 1.093]
  FRC,Scan Trimmed,Right Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Right Lower,Day 12,n=17,17 | 1.025 [0.873 to 1.204] | 1.029 [0.858 to 1.236]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19 | 1.032 [0.872 to 1.222] | 1.042 [0.924 to 1.174]
  FRC,Scan Trimmed,Left Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Left Lower,Day 12,n=17,17 | 1.012 [0.894 to 1.145] | 1.032 [0.886 to 1.201]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19 | 0.973 [0.862 to 1.097] | 1.062 [0.974 to 1.157]
  TLC,Scan Trimmed,Right Upper,Day 12,n=19,17: number analyzed (Participants) | 19 | 17
  TLC,Scan Trimmed,Right Upper,Day 12,n=19,17 | 0.991 [0.908 to 1.080] | 0.999 [0.876 to 1.141]
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,19 | 0.951 [0.870 to 1.040] | 0.964 [0.860 to 1.081]
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18 | 0.954 [0.897 to 1.014] | 0.968 [0.852 to 1.101]
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20 | 0.935 [0.860 to 1.017] | 0.950 [0.872 to 1.035]
  TLC,Scan Trimmed,Right Middle,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  TLC,Scan Trimmed,Right Middle,Day 12,n=18,17 | 0.958 [0.835 to 1.099] | 1.008 [0.891 to 1.140]
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,19 | 0.969 [0.837 to 1.122] | 0.900 [0.815 to 0.994]
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18 | 1.054 [0.936 to 1.187] | 0.963 [0.853 to 1.087]
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20 | 0.952 [0.848 to 1.068] | 0.899 [0.814 to 0.993]
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18 | 0.967 [0.911 to 1.026] | 1.004 [0.887 to 1.136]
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20 | 0.953 [0.852 to 1.066] | 0.950 [0.868 to 1.040]
  FRC,Untrimmed,Right Upper,Day 12,n= 17,16: number analyzed (Participants) | 17 | 16
  FRC,Untrimmed,Right Upper,Day 12,n= 17,16 | 0.900 [0.670 to 1.209] | 1.071 [0.851 to 1.349]
  FRC,Untrimmed,Right Upper, Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Untrimmed,Right Upper, Day 28,n=16,18 | 1.001 [0.720 to 1.390] | 1.073 [0.917 to 1.255]
  FRC,Untrimmed,Left Upper, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Left Upper, Day 12,n=18,17 | 1.001 [0.683 to 1.468] | 0.956 [0.731 to 1.251]
  Untrimmed,Left Upper, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  Untrimmed,Left Upper, Day 28,n=16,19 | 1.082 [0.669 to 1.750] | 1.065 [0.814 to 1.393]
  FRC,Untrimmed,Right Middle, Day 12,n=17,16: number analyzed (Participants) | 17 | 16
  FRC,Untrimmed,Right Middle, Day 12,n=17,16 | 1.347 [0.709 to 2.559] | 1.058 [0.825 to 1.356]
  FRC,Untrimmed,Right Middle, Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Untrimmed,Right Middle, Day 28,n=16,18 | 1.118 [0.696 to 1.797] | 1.007 [0.815 to 1.244]
  FRC,Untrimmed,Right Lower, Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Untrimmed,Right Lower, Day 12,n=17,17 | 1.237 [0.796 to 1.923] | 1.014 [0.736 to 1.397]
  FRC,Untrimmed,Right Lower, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Right Lower, Day 28,n=16,19 | 1.241 [0.841 to 1.831] | 1.031 [0.816 to 1.302]
  FRC,Untrimmed,Left Lower, Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Untrimmed,Left Lower, Day 12,n=17,17 | 0.967 [0.754 to 1.239] | 1.002 [0.702 to 1.429]
  FRC,Untrimmed,Left Lower, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Left Lower, Day 28,n=16,19 | 0.815 [0.590 to 1.125] | 1.142 [0.945 to 1.381]
  TLC,Untrimmed,Right Upper,Day 12,n=19,17: number analyzed (Participants) | 19 | 17
  TLC,Untrimmed,Right Upper,Day 12,n=19,17 | 0.982 [0.862 to 1.118] | 1.002 [0.831 to 1.209]
  TLC,Untrimmed,Right Upper, Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Untrimmed,Right Upper, Day 28,n=18,19 | 0.884 [0.776 to 1.006] | 0.941 [0.804 to 1.100]
  TLC,Untrimmed,Left Upper, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Left Upper, Day 12,n=20,18 | 0.955 [0.861 to 1.059] | 0.942 [0.789 to 1.125]
  TLC,Untrimmed,Left Upper, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Left Upper, Day 28,n=18,20 | 0.949 [0.860 to 1.046] | 0.926 [0.813 to 1.055]
  TLC,Untrimmed,Right Middle, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  TLC,Untrimmed,Right Middle, Day 12,n=18,17 | 0.942 [0.777 to 1.142] | 0.970 [0.811 to 1.161]
  TLC,Untrimmed,Right Middle, Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Untrimmed,Right Middle, Day 28,n=18,19 | 0.691 [0.475 to 1.005] | 0.892 [0.784 to 1.014]
  TLC,Untrimmed,Right Lower, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Right Lower, Day 12,n=20,18 | 1.131 [0.898 to 1.424] | 0.895 [0.745 to 1.075]
  TLC,Untrimmed,Right Lower, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Right Lower, Day 28,n=18,20 | 0.948 [0.791 to 1.135] | 0.865 [0.753 to 0.993]
  TLC,Untrimmed,Left Lower, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Left Lower, Day 12,n=20,18 | 0.982 [0.885 to 1.089] | 0.989 [0.831 to 1.178]
  TLC,Untrimmed,Left Lower, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Left Lower, Day 28,n=18,20 | 0.894 [0.693 to 1.152] | 0.967 [0.858 to 1.090]

5. Secondary Outcome: Change From Baseline (Day 12) in siVaw at FRC and TLC for Individual Lobes at Day 28
Description: siVaw is a measure of the volume in an individual's airway corrected for their lobar volume derived from the high resolution computed tomography (HRCT). It was measured at FRC and TLC. Data was collected at longitudinal time points (Untrimmed data): Baseline (Screening), Day 12 & Day 28 and at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For Untrimmed data and SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (represented by n=X1, X2 in the category title). This table presents the D12D28 scan trim pair data only.
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters per Liter
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters per Liter
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,17: number analyzed (Participants) | 16 | 17
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,17 | 0.998 [0.917 to 1.086] | 0.988 [0.909 to 1.074]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18 | 0.987 [0.905 to 1.077] | 1.014 [0.904 to 1.137]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,17: number analyzed (Participants) | 16 | 17
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,17 | 1.003 [0.876 to 1.149] | 0.930 [0.828 to 1.043]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18 | 0.938 [0.845 to 1.041] | 1.020 [0.884 to 1.176]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18 | 0.947 [0.849 to 1.057] | 1.042 [0.905 to 1.200]
  TLC, Scan Trimmed,Right Upper,Day 28,n=17,18: number analyzed (Participants) | 17 | 18
  TLC, Scan Trimmed,Right Upper,Day 28,n=17,18 | 0.963 [0.875 to 1.061] | 0.965 [0.928 to 1.004]
  TLC, Scan Trimmed,Left Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC, Scan Trimmed,Left Upper,Day 28,n=17,19 | 0.984 [0.896 to 1.079] | 0.999 [0.940 to 1.061]
  TLC, Scan Trimmed,Right Middle,Day 28,n=17,18: number analyzed (Participants) | 17 | 18
  TLC, Scan Trimmed,Right Middle,Day 28,n=17,18 | 0.807 [0.601 to 1.084] | 0.897 [0.829 to 0.971]
  TLC, Scan Trimmed,Right Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC, Scan Trimmed,Right Lower,Day 28,n=17,19 | 0.945 [0.848 to 1.052] | 0.943 [0.892 to 0.997]
  TLC, Scan Trimmed,Left Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC, Scan Trimmed,Left Lower,Day 28,n=17,19 | 0.950 [0.863 to 1.046] | 0.963 [0.868 to 1.069]

6. Secondary Outcome: Change From Baseline in siVaw at FRC and TLC for Individual Regions
Description: siVaw was measured at FRC and TLC. Data was collected at longitudinal time points (Untrimmed data): Baseline (Screening), Day 12 & Day 28 and at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For Untrimmed data and SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (n=X1, X2 in the category title).This table presents the untrimmed data (in rows with categories containing untrimmed), SCRD12 scan trim pair data (in rows with categories containing Scan Trimmed and Day 12) and SCRD28 scan trim pair data (in rows with categories containing Scan Trimmed and Day 28) only.
Time Frame: Baseline (Screening), Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters per Liter
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters per Liter
  FRC,Scan Trimmed,Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Upper,Day 12,n=18,17 | 0.996 [0.840 to 1.180] | 1.024 [0.888 to 1.181]
  FRC,Scan Trimmed,Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Upper,Day 28,n=16,19 | 1.011 [0.814 to 1.257] | 1.029 [0.934 to 1.133]
  FRC,Scan Trimmed,Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Lower,Day 12,n=17,17 | 1.003 [0.881 to 1.143] | 1.039 [0.901 to 1.199]
  FRC,Scan Trimmed,Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Lower,Day 28,n=16,19 | 0.991 [0.873 to 1.125] | 1.041 [0.942 to 1.150]
  FRC,Scan Trimmed,Central,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Central,Day 12,n=18,17 | 1.027 [0.917 to 1.151] | 1.052 [0.998 to 1.108]
  FRC,Scan Trimmed,Central,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Central,Day 28,n=16,19 | 1.048 [0.928 to 1.183] | 1.045 [0.996 to 1.096]
  FRC,Scan Trimmed,Distal,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Distal,Day 12,n=18,17 | 0.970 [0.859 to 1.096] | 1.029 [0.891 to 1.187]
  FRC,Scan Trimmed,Distal,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Distal,Day 28,n=16,19 | 0.980 [0.844 to 1.138] | 1.037 [0.945 to 1.138]
  FRC,Scan Trimmed,Total,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Total,Day 12,n=18,17 | 1.023 [0.914 to 1.144] | 1.046 [0.989 to 1.106]
  FRC,Scan Trimmed,Total,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Total,Day 28,n=16,19 | 1.041 [0.923 to 1.175] | 1.042 [0.994 to 1.091]
  TLC, Scan Trimmed,Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC, Scan Trimmed,Upper,Day 12,n=20,18 | 0.963 [0.904 to 1.026] | 0.982 [0.870 to 1.109]
  TLC, Scan Trimmed,Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC, Scan Trimmed,Upper,Day 28,n=18,20 | 0.939 [0.863 to 1.022] | 0.945 [0.865 to 1.033]
  TLC, Scan Trimmed,Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC, Scan Trimmed,Lower,Day 12,n=20,18 | 0.996 [0.924 to 1.074] | 0.982 [0.880 to 1.096]
  TLC, Scan Trimmed,Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC, Scan Trimmed,Lower,Day 28,n=18,20 | 0.958 [0.852 to 1.078] | 0.925 [0.848 to 1.009]
  TLC, Scan Trimmed,Central,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC, Scan Trimmed,Central,Day 12,n=20,18 | 1.011 [0.981 to 1.042] | 1.029 [1.000 to 1.058]
  TLC, Scan Trimmed,Central,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC, Scan Trimmed,Central,Day 28,n=18,20 | 1.013 [0.979 to 1.048] | 1.006 [0.984 to 1.028]
  TLC, Scan Trimmed,Distal,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC, Scan Trimmed,Distal,Day 12,n=20,18 | 0.979 [0.917 to 1.045] | 0.981 [0.876 to 1.098]
  TLC, Scan Trimmed,Distal,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC, Scan Trimmed,Distal,Day 28,n=18,20 | 0.948 [0.864 to 1.040] | 0.934 [0.860 to 1.015]
  TLC, Scan Trimmed,Total,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC, Scan Trimmed,Total,Day 12,n=20,18 | 1.004 [0.971 to 1.037] | 1.020 [0.982 to 1.060]
  TLC, Scan Trimmed,Total,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC, Scan Trimmed,Total,Day 28,n=18,20 | 1.001 [0.968 to 1.035] | 0.990 [0.967 to 1.014]
  FRC,Untrimmed,Upper,Day 12,n= 18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Upper,Day 12,n= 18,17 | 0.967 [0.722 to 1.296] | 1.050 [0.842 to 1.309]
  FRC,Untrimmed,Upper, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Upper, Day 28,n=16,19 | 1.027 [0.699 to 1.507] | 1.066 [0.888 to 1.279]
  FRC,Untrimmed,Lower, Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Untrimmed,Lower, Day 12,n=17,17 | 1.055 [0.786 to 1.415] | 1.026 [0.781 to 1.346]
  FRC,Untrimmed, Lower, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed, Lower, Day 28,n=16,19 | 0.991 [0.779 to 1.261] | 1.077 [0.886 to 1.308]
  FRC,Untrimmed,Central, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Central, Day 12,n=18,17 | 1.035 [0.928 to 1.153] | 1.059 [1.008 to 1.113]
  FRC,Untrimmed,Central, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Central, Day 28,n=16,19 | 1.054 [0.935 to 1.188] | 1.048 [0.994 to 1.10]
  FRC,Untrimmed,Distal, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Distal, Day 12,n=18,17 | 0.926 [0.729 to 1.177] | 1.037 [0.820 to 1.313]
  FRC,Untrimmed,Distal, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Distal, Day 28,n=16,19 | 0.981 [0.752 to 1.279] | 1.071 [0.892 to 1.285]
  FRC,Untrimmed,Total, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Total, Day 12,n=18,17 | 1.025 [0.913 to 1.151] | 1.050 [0.983 to 1.122]
  FRC,Untrimmed,Total, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Total, Day 28,n=16,19 | 1.045 [0.913 to 1.195] | 1.046 [0.988 to 1.107]
  TLC,Untrimmed,Upper,Day 12,n= 20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Upper,Day 12,n= 20,18 | 0.961 [0.853 to 1.082] | 0.959 [0.807 to 1.139]
  TLC,Untrimmed,Upper, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Upper, Day 28,n=18,20 | 0.906 [0.818 to 1.003] | 0.923 [0.815 to 1.045]
  TLC,Untrimmed,Lower, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Lower, Day 12,n=20,18 | 1.035 [0.907 to 1.182] | 0.938 [0.804 to 1.095]
  TLC,Untrimmed, Lower, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed, Lower, Day 28,n=18,20 | 0.933 [0.766 to 1.138] | 0.916 [0.820 to 1.022]
  TLC,Untrimmed,Central, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Central, Day 12,n=20,18 | 1.012 [0.985 to 1.040] | 1.027 [0.998 to 1.057]
  TLC,Untrimmed,Central, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Central, Day 28,n=18,20 | 1.010 [0.974 to 1.047] | 1.002 [0.979 to 1.026]
  TLC,Untrimmed,Distal, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Distal, Day 12,n=20,18 | 0.996 [0.882 to 1.124] | 0.946 [0.807 to 1.110]
  TLC,Untrimmed,Distal, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Distal, Day 28,n=18,20 | 0.922 [0.803 to 1.057] | 0.918 [0.824 to 1.022]
  TLC,Untrimmed,Total, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Total, Day 12,n=20,18 | 1.000 [0.970 to 1.031] | 1.009 [0.962 to 1.059]
  TLC,Untrimmed,Total, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Total, Day 28,n=18,20 | 0.993 [0.950 to 1.038] | 0.982 [0.957 to 1.008]

7. Secondary Outcome: Change From Baseline (Day 12) in siVaw at FRC and TLC for Individual Regions at Day 28
Description: as for outcome 5
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters per Liter
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters per Liter
  FRC,Scan Trimmed,Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Upper,Day 28,n=16,18 | 0.996 [0.917 to 1.082] | 0.986 [0.907 to 1.072]
  FRC,Scan Trimmed,Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Lower,Day 28,n=16,18 | 0.948 [0.862 to 1.042] | 1.025 [0.909 to 1.155]
  FRC,Scan Trimmed,Central,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Central,Day 28,n=16,18 | 0.997 [0.955 to 1.042] | 1.014 [0.955 to 1.076]
  FRC,Scan Trimmed,Distal,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Distal,Day 28,n=16,18 | 0.977 [0.898 to 1.063] | 0.996 [0.914 to 1.085]
  FRC,Scan Trimmed,Total,Day 28,n=16, 18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Total,Day 28,n=16, 18 | 0.997 [0.952 to 1.043] | 1.012 [0.953 to 1.075]
  TLC,Scan Trimmed,Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Upper,Day 28,n=17,19 | 0.973 [0.884 to 1.070] | 0.970 [0.930 to 1.012]
  TLC,Scan Trimmed,Lower,Day 28,n=17, 19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Lower,Day 28,n=17, 19 | 0.954 [0.865 to 1.051] | 0.952 [0.893 to 1.014]
  TLC,Scan Trimmed,Central,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Central,Day 28,n=17,19 | 1.009 [0.979 to 1.040] | 0.977 [0.943 to 1.012]
  TLC,Scan Trimmed,Distal,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Distal,Day 28,n=17,19 | 0.967 [0.880 to 1.063] | 0.960 [0.917 to 1.004]
  TLC,Scan Trimmed,Total,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Total,Day 28,n=17,19 | 1.003 [0.965 to 1.042] | 0.972 [0.939 to 1.006]

8. Secondary Outcome: Change From Baseline in Imaging Airway Volume (iVaw) at FRC and TLC for Individual Lobes
Description: iVaw was measured at FRC and TLC. Data was collected at longitudinal time points (Untrimmed data): Screening, Day 12 & Day 28 and at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For Untrimmed data and SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (n=X1, X2 in the category title). This table presents the untrimmed data (in rows with categories containing untrimmed), SCRD12 scan trim pair data (in rows with categories containing Scan Trimmed and Day 12) and SCRD28 scan trim pair data (in rows with categories containing Scan Trimmed and Day 28) only.
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters
  FRC,Scan Trimmed,Right Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Right Upper,Day 12,n=18,17 | 1.007 [0.847 to 1.197] | 1.044 [0.879 to 1.240]
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,19 | 1.016 [0.826 to 1.249] | 1.037 [0.931 to 1.155]
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17 | 0.965 [0.783 to 1.190] | 0.987 [0.830 to 1.173]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19 | 0.998 [0.767 to 1.299] | 1.062 [0.919 to 1.227]
  FRC,Right Middle,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Right Middle,Day 12,n=18,17 | 1.129 [0.803 to 1.588] | 1.014 [0.874 to 1.176]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,19 | 0.950 [0.739 to 1.221] | 1.018 [0.881 to 1.176]
  FRC,Right Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Right Lower,Day 12,n=17,17 | 1.046 [0.884 to 1.237] | 1.005 [0.824 to 1.225]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19 | 1.042 [0.879 to 1.235] | 1.025 [0.889 to 1.181]
  FRC,Left Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Left Lower,Day 12,n=17,17 | 1.003 [0.855 to 1.178] | 1.010 [0.832 to 1.226]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19 | 0.971 [0.836 to 1.127] | 1.029 [0.920 to 1.151]
  TLC,Scan Trimmed,Right Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Right Upper,Day 12,n=20,18 | 0.976 [0.903 to 1.054] | 0.982 [0.864 to 1.117]
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,20 | 0.941 [0.858 to 1.032] | 0.946 [0.849 to 1.054]
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18 | 0.957 [0.897 to 1.020] | 0.958 [0.840 to 1.093]
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20 | 0.928 [0.849 to 1.015] | 0.938 [0.857 to 1.025]
  TLC,Scan Trimmed,Right Middle,Day 12,n=19,18: number analyzed (Participants) | 19 | 18
  TLC,Scan Trimmed,Right Middle,Day 12,n=19,18 | 0.882 [0.810 to 0.961] | 0.988 [0.881 to 1.108]
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,20 | 0.873 [0.742 to 1.027] | 0.895 [0.811 to 0.987]
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18 | 1.083 [0.966 to 1.214] | 0.937 [0.828 to 1.061]
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20 | 0.967 [0.860 to 1.088] | 0.877 [0.782 to 0.983]
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18 | 0.981 [0.922 to 1.044] | 0.981 [0.850 to 1.131]
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20 | 0.939 [0.832 to 1.060] | 0.923 [0.843 to 1.010]
  FRC,Untrimmed,Right Upper,Day 12,n= 18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Right Upper,Day 12,n= 18,17 | 0.886 [0.652 to 1.203] | 1.095 [0.858 to 1.396]
  FRC,Untrimmed,Right Upper, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Right Upper, Day 28,n=16,19 | 0.990 [0.703 to 1.393] | 1.083 [0.923 to 1.272]
  FRC,Untrimmed,Left Upper, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Left Upper, Day 12,n=18,17 | 0.996 [0.668 to 1.485] | 0.950 [0.696 to 1.297]
  FRC,Untrimmed,Left Upper, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Left Upper, Day 28,n=16,19 | 1.071 [0.656 to 1.749] | 1.074 [0.798 to 1.444]
  FRC,Untrimmed,Right Middle, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Right Middle, Day 12,n=18,17 | 1.167 [0.633 to 2.149] | 1.157 [0.840 to 1.595]
  FRC,Untrimmed,Right Middle, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Right Middle, Day 28,n=16,19 | 0.991 [0.629 to 1.562] | 1.155 [0.819 to 1.631]
  FRC,Untrimmed,Right Lower, Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Untrimmed,Right Lower, Day 12,n=17,17 | 1.262 [0.791 to 2.015] | 0.990 [0.703 to 1.392]
  FRC,Untrimmed,Right Lower, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Right Lower, Day 28,n=16,19 | 1.253 [0.832 to 1.885] | 1.014 [0.784 to 1.311]
  FRC,Untrimmed,Left Lower, Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Untrimmed,Left Lower, Day 12,n=17,17 | 0.959 [0.714 to 1.287] | 0.981 [0.655 to 1.469]
  FRC,Untrimmed,Left Lower, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Left Lower, Day 28,n=16,19 | 0.813 [0.571 to 1.157] | 1.107 [0.882 to 1.389]
  TLC,Untrimmed,Right Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Right Upper,Day 12,n=20,18 | 0.960 [0.839 to 1.098] | 0.984 [0.822 to 1.178]
  TLC,Untrimmed,Right Upper, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Right Upper, Day 28,n=18,20 | 0.874 [0.754 to 1.012] | 0.923 [0.797 to 1.069]
  TLC,Untrimmed,Left Upper, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Left Upper, Day 12,n=20,18 | 0.958 [0.853 to 1.075] | 0.932 [0.779 to 1.116]
  TLC,Untrimmed,Left Upper, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Left Upper, Day 28,n=18,20 | 0.942 [0.850 to 1.043] | 0.914 [0.800 to 1.045]
  TLC,Untrimmed,Right Middle, Day 12,n=19,18: number analyzed (Participants) | 19 | 18
  TLC,Untrimmed,Right Middle, Day 12,n=19,18 | 0.872 [0.724 to 1.050] | 0.952 [0.806 to 1.124]
  TLC,Untrimmed,Right Middle, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Right Middle, Day 28,n=18,20 | 0.622 [0.367 to 1.053] | 0.886 [0.780 to 1.007]
  TLC,Untrimmed,Right Lower, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Right Lower, Day 12,n=20,18 | 1.162 [0.914 to 1.476] | 0.871 [0.721 to 1.053]
  TLC,Untrimmed,Right Lower, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Right Lower, Day 28,n=18,20 | 0.963 [0.795 to 1.166] | 0.843 [0.725 to 0.981]
  TLC,Untrimmed,Left Lower, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Left Lower, Day 12,n=20,18 | 0.996 [0.888 to 1.117] | 0.967 [0.797 to 1.172]
  TLC,Untrimmed,Left Lower, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Left Lower, Day 28,n=18,20 | 0.881 [0.675 to 1.149] | 0.940 [0.828 to 1.066]

9. Secondary Outcome: Change From Baseline (Day 12) in iVaw at FRC and TLC for Individual Lobes at Day 28
Description: iVaw is a measure of the volume in an individual's airway derived from the HRCT. It was measured at FRC and TLC. Data was collected at longitudinal time points (Untrimmed data): Screening, Day 12 & Day 28 and at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For Untrimmed data and SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (represented by n=X1, X2 in the category title). This table presents the D12D28 scan trim pair data only.
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18 | 0.995 [0.918 to 1.078] | 0.977 [0.880 to 1.084]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18 | 0.973 [0.891 to 1.063] | 1.016 [0.898 to 1.151]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18 | 0.958 [0.842 to 1.090] | 0.943 [0.838 to 1.061]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18 | 0.918 [0.821 to 1.025] | 1.008 [0.855 to 1.188]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18 | 0.943 [0.852 to 1.045] | 1.024 [0.877 to 1.196]
  TLC,Scan Trimmed,Right Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Right Upper,Day 28,n=17,19 | 0.963 [0.875 to 1.060] | 0.966 [0.936 to 0.997]
  TLC,Scan Trimmed,Left Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Left Upper,Day 28,n=17,19 | 0.976 [0.885 to 1.076] | 0.996 [0.942 to 1.052]
  TLC,Right Middle,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Right Middle,Day 28,n=17,19 | 0.784 [0.571 to 1.077] | 0.904 [0.841 to 0.971]
  TLC,Scan Trimmed,Right Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Right Lower,Day 28,n=17,19 | 0.926 [0.826 to 1.038] | 0.935 [0.876 to 0.997]
  TLC,Scan Trimmed,Left Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Left Lower,Day 28,n=17,19 | 0.928 [0.833 to 1.035] | 0.951 [0.855 to 1.057]

10. Secondary Outcome: Change From Baseline in iVaw at FRC and TLC for Individual Regions
Description: as for outcome 8
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters
  FRC,Scan Trimmed,Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Upper,Day 12,n=18,17 | 0.987 [0.827 to 1.178] | 1.021 [0.869 to 1.200]
  FRC,Scan Trimmed,Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Upper,Day 28,n=16,19 | 0.999 [0.800 to 1.246] | 1.039 [0.927 to 1.166]
  FRC,Scan Trimmed,Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Lower,Day 12,n=17,17 | 1.009 [0.864 to 1.178] | 1.017 [0.863 to 1.199]
  FRC,Scan Trimmed,Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Lower,Day 28,n=16,19 | 0.993 [0.862 to 1.142] | 1.018 [0.899 to 1.152]
  FRC,Scan Trimmed,Central,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Central,Day 12,n=18,17 | 1.025 [0.925 to 1.136] | 1.040 [0.985 to 1.097]
  FRC,Scan Trimmed,Central,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Central,Day 28,n=16,19 | 1.040 [0.936 to 1.155] | 1.040 [0.974 to 1.110]
  FRC,Scan Trimmed,Distal,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Distal,Day 12,n=18,17 | 0.969 [0.847 to 1.107] | 1.017 [0.866 to 1.194]
  FRC,Scan Trimmed,Distal,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Distal,Day 28,n=16,19 | 0.973 [0.834 to 1.135] | 1.032 [0.921 to 1.157]
  FRC,Scan Trimmed,Total,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Total,Day 12,n=18,17 | 1.021 [0.920 to 1.132] | 1.034 [0.970 to 1.101]
  FRC,Scan Trimmed,Total,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Total,Day 28,n=16,19 | 1.034 [0.927 to 1.153] | 1.037 [0.970 to 1.108]
  TLC,Scan Trimmed,Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Upper,Day 12,n=20,18 | 0.959 [0.899 to 1.023] | 0.973 [0.860 to 1.101]
  TLC,Scan Trimmed,Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Upper,Day 28,n=18,20 | 0.930 [0.851 to 1.015] | 0.935 [0.853 to 1.024]
  TLC,Scan Trimmed,Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Lower,Day 12,n=20,18 | 1.017 [0.945 to 1.094] | 0.960 [0.858 to 1.074]
  TLC,Scan Trimmed,Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Lower,Day 28,n=18,20 | 0.958 [0.846 to 1.084] | 0.902 [0.823 to 0.989]
  TLC,Scan Trimmed,Central,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Central,Day 12,n=20,18 | 1.019 [0.998 to 1.040] | 1.013 [0.988 to 1.040]
  TLC,Scan Trimmed,Central,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Central,Day 28,n=18,20 | 1.006 [0.984 to 1.028] | 0.989 [0.965 to 1.013]
  TLC,Scan Trimmed,Distal,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Distal,Day 12,n=20,18 | 0.986 [0.924 to 1.053] | 0.966 [0.862 to 1.083]
  TLC,Scan Trimmed,Distal,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Distal,Day 28,n=18,20 | 0.941 [0.854 to 1.038] | 0.918 [0.842 to 1.002]
  TLC,Scan Trimmed,Total,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Total,Day 12,n=20,18 | 1.011 [0.985 to 1.038] | 1.005 [0.968 to 1.043]
  TLC,Scan Trimmed,Total,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Total,Day 28,n=18,20 | 0.994 [0.967 to 1.022] | 0.973 [0.947 to 1.000]
  FRC,Untrimmed,Upper,Day 12,n= 18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Upper,Day 12,n= 18,17 | 0.959 [0.704 to 1.305] | 1.047 [0.815 to 1.345]
  FRC,Untrimmed,Upper, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Upper, Day 28,n=16,19 | 1.014 [0.685 to 1.499] | 1.076 [0.876 to 1.323]
  FRC,Untrimmed,Lower, Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Untrimmed,Lower, Day 12,n=17,17 | 1.060 [0.761 to 1.478] | 1.004 [0.741 to 1.359]
  FRC,Untrimmed, Lower, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed, Lower, Day 28,n=16,19 | 0.993 [0.750 to 1.315] | 1.052 [0.840 to 1.319]
  FRC,Untrimmed,Central, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Central, Day 12,n=18,17 | 1.033 [0.920 to 1.160] | 1.047 [0.967 to 1.134]
  FRC,Untrimmed,Central, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Central, Day 28,n=16,19 | 1.046 [0.926 to 1.182] | 1.043 [0.961 to 1.133]
  FRC,Untrimmed,Distal, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Distal, Day 12,n=18,17 | 0.924 [0.709 to 1.205] | 1.025 [0.788 to 1.333]
  FRC,Untrimmed,Distal, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Distal, Day 28,n=16,19 | 0.974 [0.735 to 1.290] | 1.066 [0.865 to 1.313]
  FRC,Untrimmed,Total, Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Untrimmed,Total, Day 12,n=18,17 | 1.023 [0.900 to 1.163] | 1.038 [0.941 to 1.145]
  FRC,Untrimmed,Total, Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Untrimmed,Total, Day 28,n=16,19 | 1.037 [0.898 to 1.198] | 1.041 [0.953 to 1.137]
  TLC,Untrimmed,Upper,Day 12,n= 20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Upper,Day 12,n= 20,18 | 0.957 [0.841 to 1.089] | 0.950 [0.800 to 1.129]
  TLC,Untrimmed,Upper, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Upper, Day 28,n=18,20 | 0.897 [0.805 to 0.998] | 0.912 [0.804 to 1.035]
  TLC,Untrimmed,Lower, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Lower, Day 12,n=20,18 | 1.057 [0.915 to 1.220] | 0.917 [0.783 to 1.074]
  TLC,Untrimmed, Lower, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed, Lower, Day 28,n=18,20 | 0.933 [0.759 to 1.147] | 0.893 [0.795 to 1.002]
  TLC,Untrimmed,Central, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Central, Day 12,n=20,18 | 1.020 [0.997 to 1.043] | 1.012 [0.984 to 1.041]
  TLC,Untrimmed,Central, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Central, Day 28,n=18,20 | 1.003 [0.976 to 1.032] | 0.985 [0.959 to 1.012]
  TLC,Untrimmed,Distal, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Distal, Day 12,n=20,18 | 1.003 [0.881 to 1.143] | 0.932 [0.795 to 1.093]
  TLC,Untrimmed,Distal, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Distal, Day 28,n=18,20 | 0.916 [0.793 to 1.056] | 0.902 [0.808 to 1.008]
  TLC,Untrimmed,Total, Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Untrimmed,Total, Day 12,n=20,18 | 1.008 [0.976 to 1.040] | 0.994 [0.949 to 1.042]
  TLC,Untrimmed,Total, Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Untrimmed,Total, Day 28,n=18,20 | 0.986 [0.945 to 1.030] | 0.965 [0.936 to 0.995]

11. Secondary Outcome: Change From Baseline (Day 12) in iVaw at FRC and TLC for Individual Regions at Day 28
Description: as for outcome 9
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Milliliters
  FRC,Scan Trimmed,Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Upper,Day 28,n=16,18 | 0.988 [0.912 to 1.070] | 0.985 [0.891 to 1.089]
  FRC,Scan Trimmed,Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Lower,Day 28,n=16,18 | 0.934 [0.847 to 1.030] | 1.010 [0.876 to 1.165]
  FRC,Scan Trimmed,Central,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Central,Day 28,n=16,18 | 0.985 [0.953 to 1.019] | 1.008 [0.942 to 1.078]
  FRC,Scan Trimmed,Distal,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Distal,Day 28,n=16,18 | 0.966 [0.891 to 1.047] | 0.990 [0.890 to 1.102]
  FRC,Scan Trimmed,Total,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Total,Day 28,n=16,18 | 0.985 [0.949 to 1.022] | 1.006 [0.938 to 1.080]
  TLC,Scan Trimmed,Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Upper,Day 28,n=17,19 | 0.968 [0.877 to 1.067] | 0.968 [0.932 to 1.005]
  TLC,Scan Trimmed,Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Lower,Day 28,n=17,19 | 0.933 [0.840 to 1.037] | 0.942 [0.879 to 1.010]
  TLC,Scan Trimmed,Central,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Central,Day 28,n=17,19 | 0.996 [0.968 to 1.024] | 0.972 [0.940 to 1.004]
  TLC,Scan Trimmed,Distal,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Distal,Day 28,n=17,19 | 0.954 [0.865 to 1.052] | 0.954 [0.912 to 0.998]
  TLC,Scan Trimmed,Total,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Total,Day 28,n=17,19 | 0.989 [0.952 to 1.028] | 0.966 [0.936 to 0.998]

12. Secondary Outcome: Change From Baseline in Imaging Airway Resistance (iRaw) at FRC and TLC for Individual Lobes
Description: iRaw is a measure of the resistance in an individual's airway derived from HRCT. It was measured at FRC and TLC. Data was collected at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (represented by n=X1, X2 in the category title). • This table presents the SCRD12 scan trim pair data (in rows with categories containing Scan Trimmed and Day 12) and SCRD28 scan trim pair data (in rows with categories containing Scan Trimmed and Day 28) only.
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Kilopascal* seconds per liter (kPa*s/L)
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Kilopascal* seconds per liter (kPa*s/L)
  FRC,Scan Trimmed,Right Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Right Upper,Day 12,n=18,17 | 1.129 [0.641 to 1.991] | 0.876 [0.477 to 1.606]
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,19 | 1.213 [0.569 to 2.586] | 0.884 [0.582 to 1.343]
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17 | 1.058 [0.631 to 1.774] | 0.951 [0.592 to 1.530]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19 | 1.151 [0.582 to 2.273] | 0.681 [0.438 to 1.060]
  FRC,Scan Trimmed,Right Middle,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Right Middle,Day 12,n=18,17 | 0.559 [0.198 to 1.576] | 0.970 [0.578 to 1.627]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,19 | 1.420 [0.573 to 3.518] | 1.275 [0.732 to 2.219]
  FRC,Scan Trimmed,Right Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Right Lower,Day 12,n=17,17 | 0.903 [0.352 to 2.314] | 1.149 [0.714 to 1.849]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19 | 0.681 [0.251 to 1.850] | 0.935 [0.512 to 1.706]
  FRC,Scan Trimmed,Left Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Left Lower,Day 12,n=17,17 | 1.084 [0.642 to 1.832] | 0.902 [0.378 to 2.157]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19 | 1.576 [0.656 to 3.785] | 0.904 [0.642 to 1.274]
  TLC,Scan Trimmed,Right Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Right Upper,Day 12,n=20,18 | 1.058 [0.820 to 1.366] | 1.057 [0.739 to 1.511]
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,20 | 1.307 [0.994 to 1.718] | 1.292 [0.951 to 1.755]
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18 | 1.129 [0.938 to 1.360] | 1.075 [0.662 to 1.747]
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20 | 1.212 [0.957 to 1.534] | 1.160 [0.851 to 1.580]
  TLC,Scan Trimmed,Right Middle,Day 12,n=19,18: number analyzed (Participants) | 19 | 18
  TLC,Scan Trimmed,Right Middle,Day 12,n=19,18 | 1.190 [0.823 to 1.720] | 1.148 [0.747 to 1.763]
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,20 | 1.749 [0.981 to 3.117] | 1.583 [1.002 to 2.502]
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18 | 0.727 [0.484 to 1.092] | 1.325 [0.860 to 2.041]
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20 | 1.143 [0.797 to 1.639] | 1.463 [1.077 to 1.988]
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18 | 1.003 [0.798 to 1.260] | 1.144 [0.714 to 1.833]
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20 | 1.259 [0.741 to 2.140] | 1.213 [0.907 to 1.623]

13. Secondary Outcome: Change From Baseline (Day 12) in iRaw at FRC and TLC for Individual Lobes at Day 28
Description: iRaw is a measure of the resistance in an individual's airway derived from HRCT. It was measured at FRC and TLC. Data was collected at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (represented by n=X1, X2 in the category title). This table presents the D12D28 scan trim pair data only.
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: kPa*s/L
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
kPa*s/L
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18 | 1.082 [0.714 to 1.641] | 1.152 [0.819 to 1.620]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18 | 1.266 [0.892 to 1.798] | 1.008 [0.641 to 1.587]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18 | 1.149 [0.709 to 1.862] | 1.477 [0.927 to 2.355]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18 | 1.269 [0.840 to 1.916] | 1.276 [0.693 to 2.350]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18 | 1.768 [0.902 to 3.465] | 1.185 [0.759 to 1.850]
  TLC,Scan Trimmed,Right Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Right Upper,Day 28,n=17,19 | 1.133 [0.798 to 1.608] | 1.143 [0.995 to 1.314]
  TLC,Scan Trimmed,Left Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Left Upper,Day 28,n=17,19 | 1.000 [0.732 to 1.367] | 1.093 [0.927 to 1.288]
  TLC,Scan Trimmed,Right Middle,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Right Middle,Day 28,n=17,19 | 1.971 [0.962 to 4.039] | 1.537 [1.055 to 2.238]
  TLC,Scan Trimmed,Right Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Right Lower,Day 28,n=17,19 | 1.408 [0.901 to 2.199] | 1.073 [0.779 to 1.478]
  TLC,Scan Trimmed,Left Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Left Lower,Day 28,n=17,19 | 1.486 [0.983 to 2.248] | 1.056 [0.691 to 1.615]

14. Secondary Outcome: Change From Baseline in iRaw at FRC and TLC for Individual Regions
Description: iRaw is a measure of the resistance in an individual's airway derived from HRCT. It was measured at FRC and TLC. Data was collected at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analyzed (n=X1, X2 in the category title). This table presents the SCRD12 scan trim pair data (in rows with categories containing Scan Trimmed and Day 12) and SCRD28 scan trim pair data (in rows with categories containing Scan Trimmed and Day 28) only.
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: kPa*s/L
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
kPa*s/L
  FRC,Scan Trimmed,Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Upper,Day 12,n=18,17 | 0.827 [0.448 to 1.526] | 0.831 [0.520 to 1.326]
  FRC,Scan Trimmed,Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Upper,Day 28,n=16,19 | 1.395 [0.682 to 2.851] | 0.776 [0.526 to 1.144]
  FRC,Scan Trimmed,Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Lower,Day 12,n=17,17 | 1.112 [0.553 to 2.236] | 1.066 [0.510 to 2.225]
  FRC,Scan Trimmed,Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Lower,Day 28,n=16,19 | 1.071 [0.515 to 2.230] | 0.912 [0.598 to 1.391]
  FRC,Scan Trimmed,Central,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Central,Day 12,n=18,17 | 0.932 [0.637 to 1.364] | 0.888 [0.729 to 1.082]
  FRC,Scan Trimmed,Central,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Central,Day 28,n=16,19 | 0.876 [0.606 to 1.266] | 0.871 [0.694 to 1.094]
  FRC,Scan Trimmed,Distal,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Distal,Day 12,n=18,17 | 1.001 [0.625 to 1.602] | 1.098 [0.563 to 2.144]
  FRC,Scan Trimmed,Distal,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Distal,Day 28,n=16,19 | 1.169 [0.559 to 2.443] | 0.857 [0.589 to 1.247]
  FRC,Scan Trimmed,Total,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Total,Day 12,n=18,17 | 0.985 [0.673 to 1.441] | 0.972 [0.711 to 1.329]
  FRC,Scan Trimmed,Total,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Total,Day 28,n=16,19 | 1.045 [0.656 to 1.665] | 0.913 [0.701 to 1.190]
  TLC,Scan Trimmed,Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Upper,Day 12,n=20,18 | 1.142 [0.888 to 1.469] | 1.167 [0.727 to 1.872]
  TLC,Scan Trimmed,Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Upper,Day 28,n=18,20 | 1.540 [1.106 to 2.145] | 1.271 [0.956 to 1.690]
  TLC,Scan Trimmed,Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Lower,Day 12,n=20,18 | 0.860 [0.649 to 1.141] | 1.206 [0.835 to 1.741]
  TLC,Scan Trimmed,Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Lower,Day 28,n=18,20 | 1.142 [0.734 to 1.775] | 1.315 [1.004 to 1.723]
  TLC,Scan Trimmed,Central,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Central,Day 12,n=20,18 | 0.987 [0.876 to 1.111] | 1.005 [0.882 to 1.146]
  TLC,Scan Trimmed,Central,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Central,Day 28,n=18,20 | 0.985 [0.914 to 1.061] | 1.057 [0.943 to 1.186]
  TLC,Scan Trimmed,Distal,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Distal,Day 12,n=20,18 | 0.959 [0.726 to 1.268] | 1.278 [0.824 to 1.983]
  TLC,Scan Trimmed,Distal,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Distal,Day 28,n=18,20 | 1.332 [0.869 to 2.040] | 1.288 [0.993 to 1.669]
  TLC,Scan Trimmed,Total,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Total,Day 12,n=20,18 | 0.993 [0.831 to 1.187] | 1.109 [0.853 to 1.443]
  TLC,Scan Trimmed,Total,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Total,Day 28,n=18,20 | 1.196 [0.959 to 1.492] | 1.202 [0.990 to 1.460]

15. Secondary Outcome: Change From Baseline (Day 12) in iRaw at FRC and TLC for Individual Regions at Day 28
Description: as for outcome 13
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: kPa*s/L
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
kPa*s/L
  FRC,Scan Trimmed,Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Upper,Day 28,n=16,18 | 1.221 [0.870 to 1.715] | 1.266 [0.848 to 1.891]
  FRC,Scan Trimmed,Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Lower,Day 28,n=16,18 | 1.531 [0.937 to 2.499] | 1.278 [0.774 to 2.112]
  FRC,Scan Trimmed,Central,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Central,Day 28,n=16,18 | 0.989 [0.873 to 1.121] | 0.926 [0.697 to 1.231]
  FRC,Scan Trimmed,Distal,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Distal,Day 28,n=16,18 | 1.373 [0.986 to 1.912] | 1.235 [0.856 to 1.781]
  FRC,Scan Trimmed,Total,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Total,Day 28,n=16,18 | 1.157 [0.940 to 1.425] | 1.001 [0.714 to 1.402]
  TLC,Scan Trimmed,Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Upper,Day 28,n=17,19 | 1.473 [0.938 to 2.313] | 1.172 [1.052 to 1.306]
  TLC,Scan Trimmed,Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Lower,Day 28,n=17,19 | 1.422 [0.942 to 2.148] | 1.089 [0.816 to 1.454]
  TLC,Scan Trimmed,Central,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Central,Day 28,n=17,19 | 0.986 [0.862 to 1.129] | 1.044 [0.937 to 1.162]
  TLC,Scan Trimmed,Distal,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Distal,Day 28,n=17,19 | 1.712 [1.119 to 2.618] | 1.079 [0.883 to 1.319]
  TLC,Scan Trimmed,Total,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Total,Day 28,n=17,19 | 1.321 [0.998 to 1.749] | 1.085 [0.933 to 1.263]

16. Secondary Outcome: Change From Baseline in Specific Imaging Airway Resistance (siRaw) at FRC and TLC for Individual Lobes
Description: siRaw is a measure of the resistance in an individual's airway corrected for their lobar volume derived from the HRCT. It was measured at FRC and TLC. Data was collected at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analysed (represented by n=X1, X2 in the category title). This table presents the SCRD12 scan trim pair data (in rows with categories containing Scan Trimmed and Day 12) and SCRD28 scan trim pair data (in rows with categories containing Scan Trimmed and Day 28) only.
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: kPa*s
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
kPa*s
  FRC,Scan Trimmed,Right Upper,Day 12,n=17,16: number analyzed (Participants) | 17 | 16
  FRC,Scan Trimmed,Right Upper,Day 12,n=17,16 | 1.117 [0.627 to 1.989] | 0.961 [0.539 to 1.711]
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,18 | 1.200 [0.574 to 2.510] | 0.923 [0.599 to 1.424]
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Left Upper,Day 12,n=18,17 | 1.053 [0.642 to 1.726] | 0.945 [0.604 to 1.479]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,19 | 1.139 [0.586 to 2.215] | 0.687 [0.457 to 1.032]
  FRC,Scan Trimmed,Right Middle,Day 12,n=17,16: number analyzed (Participants) | 17 | 16
  FRC,Scan Trimmed,Right Middle,Day 12,n=17,16 | 0.496 [0.163 to 1.511] | 1.022 [0.593 to 1.761]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,18 | 1.259 [0.521 to 3.043] | 1.424 [0.836 to 2.424]
  FRC,Scan Trimmed,Right Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Right Lower,Day 12,n=17,17 | 0.921 [0.362 to 2.342] | 1.121 [0.715 to 1.758]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,19 | 0.688 [0.257 to 1.840] | 0.920 [0.521 to 1.624]
  FRC,Scan Trimmed,Left Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Left Lower,Day 12,n=17,17 | 1.075 [0.648 to 1.785] | 0.884 [0.386 to 2.021]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,19 | 1.573 [0.669 to 3.701] | 0.876 [0.634 to 1.212]
  TLC,Scan Trimmed,Right Upper,Day 12,n=19,17: number analyzed (Participants) | 19 | 17
  TLC,Scan Trimmed,Right Upper,Day 12,n=19,17 | 1.037 [0.788 to 1.364] | 1.035 [0.711 to 1.509]
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Scan Trimmed,Right Upper,Day 28,n=18,19 | 1.292 [0.992 to 1.684] | 1.262 [0.912 to 1.747]
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Upper,Day 12,n=20,18 | 1.133 [0.946 to 1.358] | 1.064 [0.659 to 1.720]
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Upper,Day 28,n=18,20 | 1.203 [0.955 to 1.515] | 1.145 [0.843 to 1.554]
  TLC,Scan Trimmed,Right Middle,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  TLC,Scan Trimmed,Right Middle,Day 12,n=18,17 | 1.094 [0.730 to 1.639] | 1.101 [0.690 to 1.758]
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Scan Trimmed,Right Middle,Day 28,n=18,19 | 1.575 [0.965 to 2.570] | 1.557 [0.955 to 2.538]
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Right Lower,Day 12,n=20,18 | 0.747 [0.498 to 1.120] | 1.290 [0.842 to 1.976]
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Right Lower,Day 28,n=18,20 | 1.161 [0.814 to 1.654] | 1.427 [1.065 to 1.912]
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Left Lower,Day 12,n=20,18 | 1.018 [0.810 to 1.278] | 1.118 [0.715 to 1.747]
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Left Lower,Day 28,n=18,20 | 1.240 [0.735 to 2.092] | 1.178 [0.876 to 1.584]

17. Secondary Outcome: Change From Baseline (Day 12) in Specific Imaging Airway Resistance (siRaw) at FRC and TLC for Individual Lobes at Day 28
Description: siRaw is a measure of the resistance in an individual's airway corrected for their lobar volume derived from the HRCT. It was measured at FRC and TLC. Data was collected at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe) and 5 Regions (Upper, Lower, Central, Distal & Total). For SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only participants available at the specified time point were analysed (represented by n=X1, X2 in the category title). This table presents the D12D28 scan trim pair data only.
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: kPa*s
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
kPa*s
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,17: number analyzed (Participants) | 16 | 17
  FRC,Scan Trimmed,Right Upper,Day 28,n=16,17 | 1.079 [0.711 to 1.636] | 1.073 [0.794 to 1.451]
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Upper,Day 28,n=16,18 | 1.249 [0.886 to 1.760] | 1.011 [0.653 to 1.566]
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,17: number analyzed (Participants) | 16 | 17
  FRC,Scan Trimmed,Right Middle,Day 28,n=16,17 | 1.097 [0.647 to 1.859] | 1.354 [0.885 to 2.070]
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Right Lower,Day 28,n=16,18 | 1.241 [0.845 to 1.822] | 1.261 [0.706 to 2.252]
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Left Lower,Day 28,n=16,18 | 1.760 [0.893 to 3.470] | 1.165 [0.755 to 1.798]
  TLC,Scan Trimmed,Right Upper,Day 28,n=17,18: number analyzed (Participants) | 17 | 18
  TLC,Scan Trimmed,Right Upper,Day 28,n=17,18 | 1.132 [0.796 to 1.611] | 1.142 [0.977 to 1.336]
  TLC,Scan Trimmed,Left Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Left Upper,Day 28,n=17,19 | 0.992 [0.730 to 1.349] | 1.089 [0.921 to 1.288]
  TLC,Scan Trimmed,Right Middle,Day 28,n=17,18: number analyzed (Participants) | 17 | 18
  TLC,Scan Trimmed,Right Middle,Day 28,n=17,18 | 1.915 [0.956 to 3.834] | 1.564 [1.042 to 2.347]
  TLC,Scan Trimmed,Right Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Right Lower,Day 28,n=17,19 | 1.380 [0.894 to 2.130] | 1.064 [0.783 to 1.447]
  TLC,Scan Trimmed,Left Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Left Lower,Day 28,n=17,19 | 1.453 [0.977 to 2.161] | 1.042 [0.683 to 1.590]

18. Secondary Outcome: Change From Baseline in Specific Imaging Airway Resistance (siRaw) at FRC and TLC for Individual Regions
Description: as for outcome 16
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: kPa*s
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
kPa*s
  FRC,Scan Trimmed,Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Upper,Day 12,n=18,17 | 0.820 [0.443 to 1.517] | 0.828 [0.531 to 1.292]
  FRC,Scan Trimmed,Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Upper,Day 28,n=16,19 | 1.377 [0.679 to 2.793] | 0.784 [0.546 to 1.124]
  FRC,Scan Trimmed,Lower,Day 12,n=17,17: number analyzed (Participants) | 17 | 17
  FRC,Scan Trimmed,Lower,Day 12,n=17,17 | 1.118 [0.559 to 2.239] | 1.043 [0.516 to 2.109]
  FRC,Scan Trimmed,Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Lower,Day 28,n=16,19 | 1.073 [0.529 to 2.177] | 0.891 [0.601 to 1.321]
  FRC,Scan Trimmed,Central,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Central,Day 12,n=18,17 | 0.931 [0.634 to 1.367] | 0.878 [0.734 to 1.050]
  FRC,Scan Trimmed,Central,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Central,Day 28,n=16,19 | 0.870 [0.598 to 1.265] | 0.867 [0.709 to 1.060]
  FRC,Scan Trimmed,Distal,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Distal,Day 12,n=18,17 | 0.999 [0.617 to 1.617] | 1.085 [0.567 to 2.077]
  FRC,Scan Trimmed,Distal,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Distal,Day 28,n=16,19 | 1.161 [0.566 to 2.380] | 0.853 [0.604 to 1.204]
  FRC,Scan Trimmed,Total,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Scan Trimmed,Total,Day 12,n=18,17 | 0.983 [0.674 to 1.435] | 0.961 [0.717 to 1.287]
  FRC,Scan Trimmed,Total,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Scan Trimmed,Total,Day 28,n=16,19 | 1.038 [0.656 to 1.641] | 0.909 [0.719 to 1.150]
  TLC,Scan Trimmed,Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Upper,Day 12,n=20,18 | 1.139 [0.886 to 1.464] | 1.156 [0.723 to 1.849]
  TLC,Scan Trimmed,Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Upper,Day 28,n=18,20 | 1.524 [1.101 to 2.111] | 1.257 [0.950 to 1.664]
  TLC,Scan Trimmed,Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Lower,Day 12,n=20,18 | 0.878 [0.665 to 1.161] | 1.179 [0.822 to 1.690]
  TLC,Scan Trimmed,Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Lower,Day 28,n=18,20 | 1.142 [0.740 to 1.760] | 1.282 [0.982 to 1.673]
  TLC,Scan Trimmed,Central,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Central,Day 12,n=20,18 | 0.994 [0.883 to 1.120] | 0.990 [0.870 to 1.127]
  TLC,Scan Trimmed,Central,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Central,Day 28,n=18,20 | 0.978 [0.904 to 1.059] | 1.039 [0.931 to 1.160]
  TLC,Scan Trimmed,Distal,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Distal,Day 12,n=20,18 | 0.966 [0.735 to 1.271] | 1.259 [0.815 to 1.946]
  TLC,Scan Trimmed,Distal,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Distal,Day 28,n=18,20 | 1.323 [0.869 to 2.014] | 1.266 [0.981 to 1.633]
  TLC,Scan Trimmed,Total,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Scan Trimmed,Total,Day 12,n=20,18 | 1.000 [0.840 to 1.191] | 1.093 [0.844 to 1.416]
  TLC,Scan Trimmed,Total,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Scan Trimmed,Total,Day 28,n=18,20 | 1.188 [0.958 to 1.473] | 1.181 [0.978 to 1.427]

19. Secondary Outcome: Change From Baseline (Day 12) in Specific Imaging Airway Resistance (siRaw) at FRC and TLC for Individual Regions at Day 28
Description: as for outcome 17
Time Frame: Baseline (Day 12) and Day 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: kPa*s
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
kPa*s
  FRC,Scan Trimmed,Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Upper,Day 28,n=16,18 | 1.211 [0.852 to 1.722] | 1.265 [0.872 to 1.836]
  FRC,Scan Trimmed,Lower,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Lower,Day 28,n=16,18 | 1.508 [0.929 to 2.448] | 1.260 [0.778 to 2.041]
  FRC,Scan Trimmed,Central,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Central,Day 28,n=16,18 | 0.977 [0.861 to 1.110] | 0.921 [0.703 to 1.206]
  FRC,Scan Trimmed,Distal,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Distal,Day 28,n=16,18 | 1.356 [0.980 to 1.877] | 1.227 [0.876 to 1.720]
  FRC,Scan Trimmed,Total,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Scan Trimmed,Total,Day 28,n=16,18 | 1.144 [0.922 to 1.418] | 0.995 [0.723 to 1.368]
  TLC,Scan Trimmed,Upper,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Upper,Day 28,n=17,19 | 1.465 [0.934 to 2.300] | 1.169 [1.050 to 1.302]
  TLC,Scan Trimmed,Lower,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Lower,Day 28,n=17,19 | 1.392 [0.936 to 2.072] | 1.079 [0.813 to 1.430]
  TLC,Scan Trimmed,Central,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Central,Day 28,n=17,19 | 0.973 [0.853 to 1.111] | 1.038 [0.935 to 1.153]
  TLC,Scan Trimmed,Distal,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Distal,Day 28,n=17,19 | 1.689 [1.111 to 2.567] | 1.073 [0.882 to 1.305]
  TLC,Scan Trimmed,Total,Day 28,n=17,19: number analyzed (Participants) | 17 | 19
  TLC,Scan Trimmed,Total,Day 28,n=17,19 | 1.303 [0.990 to 1.717] | 1.079 [0.932 to 1.250]

20. Secondary Outcome: Change From Baseline in Lung Lobar Volume (iVlobe) at FRC and TLC for Individual Lobes
Description: Change from Baseline in lung lobar volumes was measured at FRC and TLC scan conditions. Data was collected at longitudinal time points: Baseline (Screening), Day 12 and Day 28. At each time point it was measure at 5 lobes (right upper lobe, left upper lobe, right middle lobe, right lower lobe & left lower lobe). The value at Screening was considered as Baseline. Change from baseline is the post-Baseline value minus the Baseline value. The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI.There was no intent to compare two devices.
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Liters
  FRC,Right Upper,Day 12,n=17,16: number analyzed (Participants) | 17 | 16
  FRC,Right Upper,Day 12,n=17,16 | 0.989 [0.921 to 1.063] | 0.971 [0.935 to 1.009]
  FRC,Right Upper,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Right Upper,Day 28,n=16,18 | 0.989 [0.929 to 1.053] | 0.999 [0.952 to 1.048]
  FRC,Left Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Left Upper,Day 12,n=18,17 | 0.995 [0.938 to 1.056] | 0.993 [0.924 to 1.068]
  FRC,Left Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Left Upper,Day 28,n=16,19 | 0.990 [0.935 to 1.048] | 1.008 [0.955 to 1.064]
  FRC,Right Middle,Day 12,n=17,16: number analyzed (Participants) | 17 | 16
  FRC,Right Middle,Day 12,n=17,16 | 0.931 [0.819 to 1.057] | 0.979 [0.949 to 1.010]
  FRC,Right Middle,Day 28,n=16,18: number analyzed (Participants) | 16 | 18
  FRC,Right Middle,Day 28,n=16,18 | 0.887 [0.708 to 1.111] | 1.010 [0.964 to 1.060]
  FRC,Right Lower,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Right Lower,Day 12,n=18,17 | 1.021 [0.928 to 1.123] | 0.976 [0.908 to 1.048]
  FRC,Right Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Right Lower,Day 28,n=16,19 | 1.009 [0.907 to 1.124] | 0.984 [0.927 to 1.044]
  FRC,Left Lower,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Left Lower,Day 12,n=18,17 | 0.996 [0.917 to 1.082] | 0.979 [0.905 to 1.059]
  FRC,Left Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Left Lower,Day 28,n=16,19 | 0.998 [0.915 to 1.089] | 0.969 [0.898 to 1.045]
  TLC,Right Upper,Day 12,n=19,17: number analyzed (Participants) | 19 | 17
  TLC,Right Upper,Day 12,n=19,17 | 0.991 [0.964 to 1.020] | 0.992 [0.976 to 1.007]
  TLC,Right Upper,Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Right Upper,Day 28,n=18,19 | 0.989 [0.967 to 1.012] | 0.984 [0.965 to 1.004]
  TLC,Left Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Left Upper,Day 12,n=20,18 | 1.003 [0.985 to 1.022] | 0.990 [0.975 to 1.005]
  TLC,Left Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Left Upper,Day 28,n=18,20 | 0.992 [0.978 to 1.008] | 0.987 [0.968 to 1.006]
  TLC,Right Middle,Day 12,n=19,17: number analyzed (Participants) | 19 | 17
  TLC,Right Middle,Day 12,n=19,17 | 0.935 [0.815 to 1.072] | 0.990 [0.960 to 1.022]
  TLC,Right Middle,Day 28,n=18,19: number analyzed (Participants) | 18 | 19
  TLC,Right Middle,Day 28,n=18,19 | 0.900 [0.741 to 1.094] | 0.998 [0.969 to 1.028]
  TLC,Right Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Right Lower,Day 12,n=20,18 | 1.027 [0.981 to 1.076] | 0.973 [0.950 to 0.997]
  TLC,Right Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Right Lower,Day 28,n=18,20 | 1.016 [0.963 to 1.072] | 0.975 [0.946 to 1.005]
  TLC,Left Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Left Lower,Day 12,n=20,18 | 1.015 [0.982 to 1.048] | 0.977 [0.937 to 1.019]
  TLC,Left Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Left Lower,Day 28,n=18,20 | 0.985 [0.953 to 1.018] | 0.971 [0.929 to 1.015]

21. Secondary Outcome: Change From Baseline in Lung Lobar Volume (iVlobe) at FRC and TLC for Individual Regions
Description: Change from Baseline in lung lobar volumes was measured at FRC and TLC scan conditions. Data was collected at longitudinal time points: Baseline (Screening), Day 12 and Day 28. At each time point it was measure at 5 Regions (Upper, Lower, Central, Distal & Total). The value at Screening was considered as Baseline. Change from Baseline is the post-Baseline value minus the Baseline value. The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI.There was no intent to compare two devices.
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Liters
  FRC,Upper,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Upper,Day 12,n=18,17 | 0.991 [0.935 to 1.051] | 0.997 [0.932 to 1.068]
  FRC,Upper,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Upper,Day 28,n=16,19 | 0.987 [0.932 to 1.045] | 1.010 [0.961 to 1.061]
  FRC,Lower,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Lower,Day 12,n=18,17 | 1.008 [0.923 to 1.100] | 0.979 [0.911 to 1.051]
  FRC,Lower,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Lower,Day 28,n=16,19 | 1.002 [0.912 to 1.101] | 0.978 [0.918 to 1.041]
  FRC,Total,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Total,Day 12,n=18,17 | 0.998 [0.931 to 1.070] | 0.988 [0.925 to 1.056]
  FRC,Total,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Total,Day 28,n=16,19 | 0.993 [0.925 to 1.065] | 0.995 [0.944 to 1.049]
  TLC,Upper,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Upper,Day 12,n=20,18 | 0.997 [0.980 to 1.013] | 0.991 [0.978 to 1.004]
  TLC,Upper,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Upper,Day 28,n=18,20 | 0.990 [0.978 to 1.002] | 0.989 [0.972 to 1.006]
  TLC,Lower,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Lower,Day 12,n=20,18 | 1.021 [0.985 to 1.057] | 0.977 [0.954 to 1.001]
  TLC,Lower,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Lower,Day 28,n=18,20 | 1.000 [0.961 to 1.040] | 0.975 [0.947 to 1.004]
  TLC,Total,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Total,Day 12,n=20,18 | 1.008 [0.985 to 1.030] | 0.985 [0.970 to 1.000]
  TLC,Total,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Total,Day 28,n=18,20 | 0.993 [0.972 to 1.015] | 0.983 [0.962 to 1.004]

22. Secondary Outcome: Change From Baseline in Trachea Length and Diameter at FRC and TLC
Description: Trachea length and diameter was derived from HRCT. It was measured at both FRC and TLC scan conditions. The value at Screening was considered as Baseline. Change from Baseline is the post-Baseline value minus the Baseline value. The change from Baseline data is presented for Day 12 and Day 28 for trachea length and diameter. The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI.There was no intent to compare two devices.
Time Frame: Baseline (Screening) and Days 12 and 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimeters
Groups:
- All NEMI: Participants were administered with placebo matching NEMI once daily in the morning before breakfast for 84 consecutive days using DISKUS or ELLIPTA dry powder inhaler (DPI).
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Millimeters
  FRC,Length,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Length,Day 12,n=18,17 | 0.094 (7.2507) | 0.972 (6.5552)
  FRC,Length,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Length,Day 28,n=16,19 | 0.796 (7.7795) | 0.281 (5.1808)
  FRC,Diameter,Day 12,n=18,17: number analyzed (Participants) | 18 | 17
  FRC,Diameter,Day 12,n=18,17 | 0.225 (1.3641) | 0.252 (1.0023)
  FRC,Diameter,Day 28,n=16,19: number analyzed (Participants) | 16 | 19
  FRC,Diameter,Day 28,n=16,19 | 0.225 (1.3812) | 0.116 (1.1600)
  TLC,Length,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Length,Day 12,n=20,18 | -0.164 (2.8331) | 0.827 (3.1842)
  TLC,Length,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Length,Day 28,n=18,20 | -0.094 (2.8480) | 0.069 (3.4882)
  TLC,Diameter,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  TLC,Diameter,Day 12,n=20,18 | 0.134 (0.4670) | 0.070 (0.4222)
  TLC,Diameter,Day 28,n=18,20: number analyzed (Participants) | 18 | 20
  TLC,Diameter,Day 28,n=18,20 | 0.076 (0.4751) | -0.188 (0.4983)

23. Secondary Outcome: Change From Baseline (Average Day 1 to 3) Peak Expiratory Flow (PEF)
Description: PEF measurements were taken (in triplicate) daily in the morning before dose administration, as soon as it is safe for the participant to do so. The best/highest result was recorded. Participants were provided with a handheld device. Baseline here is defined as average of Day 1 to Day 3. Change from Baseline is the post-Baseline value minus the Baseline value. The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI. There was no intent to compare two devices.
Time Frame: Baseline and up to Day 84
Population: All Subjects Population.
Measure: Mean (95% Confidence Interval); unit: Liters per minute
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Liters per minute
  Day 4 | 2.5 [-3.0 to 11.4] | 4.1 [-5.4 to 13.7]
  Day 5 | -3.0 [-12.8 to 6.8] | 6.3 [-4.1 to 16.8]
  Day 6 | 7.3 [-3.7 to 18.4] | 7.5 [-6.2 to 21.3]
  Day 7 | 8.1 [-3.0 to 19.3] | 11.3 [-1.3 to 24.0]
  Day 8 | 0.8 [-12.7 to 14.4] | 8.2 [-5.3 to 21.8]
  Day 9 | 10.0 [-5.5 to 25.7] | 17.7 [-1.4 to 37.0]
  Day 10 | 12.9 [-2.2 to 28.2] | 15.2 [2.8 to 27.6]
  Day 11 | 14.1 [-3.3 to 31.5] | 21.1 [1.2 to 41.0]
  Day 12 | 6.2 [-11.2 to 23.8] | 20.4 [2.2 to 38.7]
  Day 13 | 21.0 [-4.5 to 46.6] | 18.8 [-3.1 to 40.8]
  Day 14 | 9.4 [-11.7 to 30.7] | 15.3 [-0.2 to 30.8]
  Day 15 | 17.7 [-2.3 to 37.7] | 10.8 [-6.2 to 28.0]
  Day 16 | 14.1 [-10.7 to 39.0] | 12.5 [-1.8 to 26.8]
  Day 17 | 17.6 [-3.9 to 39.3] | 11.5 [-1.7 to 24.7]
  Day 18 | 11.8 [-10.6 to 34.3] | 11.9 [-3.7 to 27.5]
  Day 19 | 12.9 [-4.1 to 30.1] | 7.1 [-7.2 to 21.5]
  Day 20 | 6.4 [-16.5 to 29.4] | 3.3 [-9.3 to 16.0]
  Day 21 | 20.1 [4.5 to 35.6] | 4.1 [-7.8 to 16.1]
  Day 22 | 10.7 [-11.0 to 32.5] | 6.2 [-5.0 to 17.6]
  Day 23 | 16.0 [-5.2 to 37.3] | 2.8 [-7.3 to 13.1]
  Day 24 | 19.0 [-5.3 to 43.5] | 6.9 [-7.6 to 21.4]
  Day 25 | 23.8 [2.9 to 44.7] | 11.6 [-2.8 to 26.1]
  Day 26 | 20.8 [0.8 to 40.7] | 14.4 [-0.9 to 29.7]
  Day 27 | 29.1 [3.8 to 54.5] | 17.6 [-5.4 to 40.7]
  Day 28 | 19.3 [-2.7 to 41.4] | 11.2 [-7.9 to 30.4]
  Day 29 | 20.8 [-3.5 to 45.2] | 13.8 [-6.4 to 34.2]
  Day 30 | 9.5 [-16.2 to 35.3] | 17.2 [-7.2 to 41.7]
  Day 31 | 9.5 [-11.9 to 31.0] | 11.5 [-8.1 to 31.1]
  Day 32 | 5.9 [-18.7 to 30.5] | 17.2 [-1.9 to 36.4]
  Day 33 | 9.5 [-15.2 to 34.3] | 7.3 [-15.7 to 30.3]
  Day 34 | 6.4 [-22.3 to 35.3] | 6 [-5.0 to 17.0]
  Day 35 | 17.0 [-6.0 to 40.1] | 7 [-3.5 to 17.5]
  Day 36 | 16.7 [-4.2 to 37.7] | 3 [-9.0 to 15.0]
  Day 37 | 13.4 [-8.4 to 35.2] | 9.2 [-1.9 to 20.4]
  Day 38 | 12.6 [-7.4 to 32.6] | 5.5 [-5.9 to 16.9]
  Day 39 | 13.4 [-8.1 to 35.0] | 9.5 [-6.4 to 25.4]
  Day 40 | 13.7 [-8.6 to 36.0] | 10 [-5.1 to 25.1]
  Day 41 | 16.7 [-10.1 to 43.6] | 8 [-7.6 to 23.6]
  Day 42 | 16.7 [-8.2 to 41.7] | 10.2 [-6.3 to 26.8]
  Day 43 | 16.4 [-5.8 to 38.8] | 15 [-1.0 to 31.0]
  Day 44 | 12.6 [-14.2 to 39.4] | 9.5 [-5.33 to 24.3]
  Day 45 | 14.5 [-7.0 to 36.1] | 7.5 [-5.8 to 20.8]
  Day 46 | 9.7 [-8.8 to 28.2] | 5 [-9.2 to 19.2]
  Day 47 | 12.3 [-6.4 to 31.1] | 7.2 [-6.9 to 21.4]
  Day 48 | 13.4 [-13.1 to 40.0] | 6.2 [-9.7 to 22.2]
  Day 49 | 14.5 [-11.1 to 40.2] | 12.8 [-3.3 to 28.9]
  Day 50 | 20.1 [-0.5 to 40.7] | 9.7 [-7.5 to 27.0]
  Day 51 | 18.9 [-4.8 to 42.7] | 13.2 [-6.9 to 33.4]
  Day 52 | 14.5 [-7.3 to 36.4] | 21.5 [0.1 to 43.0]
  Day 53 | 8.9 [-11.9 to 29.9] | 17.3 [-4.6 to 39.3]
  Day 54 | 10.6 [-10.8 to 32.1] | 14.4 [-4.3 to 33.2]
  Day 55 | 21.0 [-14.4 to 56.6] | 18.7 [-5.4 to 43.0]
  Day 56 | 12.5 [-11.1 to 36.2] | 26.5 [-0.3 to 53.4]
  Day 57 | 16.2 [-6.8 to 39.3] | 32.3 [5.9 to 58.7]
  Day 58 | 14.2 [-9.3 to 37.8] | 10.4 [-7.2 to 28.1]
  Day 59 | 15.1 [-7.9 to 38.1] | 11.2 [-2.84 to 25.3]
  Day 60 | 16.4 [-12.5 to 45.5] | 1.2 [-11.1 to 13.6]
  Day 61 | 18.9 [-1.9 to 39.9] | 5.7 [-9.0 to 20.5]
  Day 62 | 16.9 [-6.5 to 40.4] | 10.2 [-6.6 to 27.1]
  Day 63 | 22.4 [-2.7 to 47.6] | 7.2 [-8.6 to 23.1]
  Day 64 | 7.9 [-16.0 to 31.9] | 9.5 [-5.9 to 24.9]
  Day 65 | 12.9 [-4.9 to 30.9] | 15 [-3.7 to 33.7]
  Day 66 | 10.0 [-9.2 to 29.4] | 10 [-5.3 to 25.3]
  Day 67 | 12.7 [-7.2 to 32.7] | 15.2 [-4.4 to 34.9]
  Day 68 | 14.3 [-5.0 to 33.6] | 11 [-4.02 to 26.0]
  Day 69 | 11.9 [-5.6 to 29.5] | 11.5 [-6.0 to 29.0]
  Day 70 | 10.8 [-6.4 to 28.2] | 11.2 [-4.0 to 26.5]
  Day 71 | 7.9 [-11.0 to 26.9] | 11 [-5.31 to 27.3]
  Day 72 | 7.9 [-11.3 to 27.2] | 14.9 [-0.3 to 30.1]
  Day 73 | 3.2 [-8.2 to 14.7] | 14.3 [-5.3 to 34.0]
  Day 74 | 6.2 [-10.0 to 22.6] | 10.7 [-6.7 to 28.2]
  Day 75 | 7.13 [-10.3 to 24.6] | 13 [-7.4 to 33.4]
  Day 76 | 12.1 [-6.4 to 30.7] | 11.2 [-8.2 to 30.7]
  Day 77 | 12.3 [-15.6 to 40.2] | 16.5 [-5.1 to 38.1]
  Day 78 | 10.4 [-9.9 to 30.8] | 12 [-4.2 to 28.2]
  Day 79 | 21.2 [-5.9 to 48.4] | 9.7 [-10.3 to 29.8]
  Day 80 | 18.1 [-7.1 to 43.3] | 10 [-8.0 to 28.0]
  Day 81 | 7.3 [-8.6 to 23.2] | 7 [-11.0 to 25.0]
  Day 82 | 5.6 [-11.5 to 22.8] | 10 [-7.2 to 27.2]
  Day 83 | 21.1 [-7.7 to 49.9] | 13.0 [-5.7 to 31.8]
  Day 84 | 12.9 [-14.9 to 40.9] | 11.6 [-19.7 to 43.0]

24. Secondary Outcome: Mean Number of Occasions of Rescue Usage Per Day
Description: For reliever/rescue use, bronchodilator use recorded in the diary was summarized as the mean number of occasions of rescue use per day.where a rescue-free day was defined as a 24-hour period in which the number of occasions of bronchodilator use was zero. Number of occasions bronchodilator taken in the last 24 hours were collected in the daily diary. The mean number of occasions of rescue use per day, were calculated for each participant during the four weekly periods (Weeks 1 to 4; Weeks 5-8 and Weeks 9-12). The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI.There was no intent to compare two devices.
Time Frame: Weeks 1 to 4; Weeks 5 to 8 and Weeks 9 to 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Rescue use per day
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Rescue use per day
  Weeks 1-4,n=22,21: number analyzed (Participants) | 22 | 21
  Weeks 1-4,n=22,21 | 3.05 (2.520) | 2.77 (2.432)
  Weeks 5-8,n=19,20: number analyzed (Participants) | 19 | 20
  Weeks 5-8,n=19,20 | 2.93 (2.342) | 2.81 (2.827)
  Weeks 9-12,n=19,20: number analyzed (Participants) | 19 | 20
  Weeks 9-12,n=19,20 | 3.19 (2.065) | 2.84 (2.569)

25. Secondary Outcome: Mean Rescue Medication Free Days
Description: For reliever/rescue use, bronchodilator use recorded in the diary was summarized as the mean number of occasions of rescue use per day, where a rescue-free day was defined as a 24-hour period in which the number of occasions of bronchodilator use was zero. Number of occasions bronchodilator taken in the last 24 hours were collected in the daily diary. The mean number of rescue free days were calculated for each participant during the four weekly periods (Weeks 1 to 4; Weeks 5-8 and Weeks 9-12). The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI. There was no intent to compare two devices.
Time Frame: Weeks 1 to 4; Weeks 5 to 8 and Weeks 9 to 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Days
  Weeks 1-4,n=22,21: number analyzed (Participants) | 22 | 21
  Weeks 1-4,n=22,21 | 7.5 (9.21) | 7.7 (10.06)
  Weeks 5-8,n=19,20: number analyzed (Participants) | 19 | 20
  Weeks 5-8,n=19,20 | 5.8 (8.58) | 9.0 (12.14)
  Weeks 9-12,n=19,20: number analyzed (Participants) | 19 | 20
  Weeks 9-12,n=19,20 | 3.7 (6.68) | 7.9 (11.14)

26. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC)
Description: FEV1 is the volume of air that can forcibly be blown out in one second. A triplicate FEV1 measurement were taken daily in the morning before dose administration using the site's spirometer as soon as it was safe to do so. FVC is defined as the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. Baseline is the latest available measurement from Day 2 Within 48 hours /discharge (On Treatment) and Day 1 (Pre-Treatment). Change from Baseline is the post-Baseline value minus Baseline value. The study had a protocol amendment to reflect changes in manufacturing device from DISKUS to ELLIPTA after study had been initiated, but the 2 treatment arms remained the same i.e. Placebo and NEMI.There was no intent to compare two devices.
Time Frame: Baseline and Days 12, 28, 56, 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | All Placebo | All NEMI
Number analyzed (Participants) | 22 | 22
Liters
  FEV1,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  FEV1,Day 12,n=20,18 | -0.001 (0.1681) | 0.084 (0.1879)
  FEV1,Day 28,n=19,20: number analyzed (Participants) | 19 | 20
  FEV1,Day 28,n=19,20 | 0.005 (0.2227) | 0.094 (0.2035)
  FEV1,Day 56,n=19,20: number analyzed (Participants) | 19 | 20
  FEV1,Day 56,n=19,20 | -0.014 (0.1783) | 0.112 (0.2613)
  FEV1,Day 84,n=17,20: number analyzed (Participants) | 17 | 20
  FEV1,Day 84,n=17,20 | -0.029 (0.1281) | 0.077 (0.2747)
  FVC,Day 12,n=20,18: number analyzed (Participants) | 20 | 18
  FVC,Day 12,n=20,18 | -0.024 (0.4723) | 0.062 (0.3770)
  FVC,Day 28,n=19,20: number analyzed (Participants) | 19 | 20
  FVC,Day 28,n=19,20 | 0.024 (0.4159) | 0.231 (0.4270)
  FVC,Day 56,n=19,20: number analyzed (Participants) | 19 | 20
  FVC,Day 56,n=19,20 | -0.078 (0.4106) | 0.212 (0.4827)
  FVC,Day 84,n=17,20: number analyzed (Participants) | 17 | 20
  FVC,Day 84,n=17,20 | -0.104 (0.3786) | 0.123 (0.4579)

27. Secondary Outcome: Number of Participants With Worst Case Hematology Results Post-Baseline Relative to Baseline
Description: Blood samples were collected to analyze the following s hematology parameters: Hemoglobin, Hematocrit, Mean Corpuscle Hemoglobin (MCH), Mean Corpuscle Volume (MCV), Platelet count, Red Blood Cell (RBC) count, White Blood Cell (WBC) count, Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils. Participants were counted in the worst case category that their value changes to (low or high), unless there is no change in their category. Participants whose lab value category was unchanged (example given [e.g.],High to High), or whose value became normal, were not recorded. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. The value at Screening was considered as Baseline. Data for Worst Case Laboratory Hematology values Post-Baseline Relative to Baseline has been presented.
Time Frame: Baseline (Screening) and up to 14 weeks
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Via DISKUS: Participants were administered with placebo matching NEMI once daily in the morning before breakfast for 84 consecutive days using DISKUS DPI.
- NEMI 1000 mcg Via DISKUS: Participants were administered with NEMI 1000 mcg once daily in the morning before breakfast for 84 consecutive days using DISKUS DPI.
- Placebo Via ELLIPTA: Participants were administered with placebo matching NEMI once daily in the morning before breakfast for 84 consecutive days using ELLIPTA DPI.
- NEMI 700 mcg Via ELLIPTA: Participants were administered with NEMI 700 mcg once daily in the morning before breakfast for 84 consecutive days using ELLIPTA DPI.
Arm/Group | Placebo Via DISKUS | NEMI 1000 mcg Via DISKUS | Placebo Via ELLIPTA | NEMI 700 mcg Via ELLIPTA
Number analyzed (Participants) | 14 | 14 | 8 | 8
Participants
  Basophils,To Low | 0 | 0 | 0 | 0
  Basophils,To High | 0 | 0 | 0 | 0
  Eosinophils,To Low | 2 | 4 | 1 | 0
  Eosinophils,To High | 1 | 1 | 0 | 1
  Hemoglobin,To Low | 0 | 0 | 0 | 0
  Hemoglobin,To High | 1 | 0 | 0 | 2
  Hematocrit,To Low | 0 | 0 | 0 | 0
  Hematocrit,To High | 3 | 3 | 0 | 0
  Lymphocytes,To Low | 0 | 1 | 0 | 1
  Lymphocytes,To High | 1 | 0 | 0 | 0
  MCH,To Low | 0 | 1 | 0 | 0
  MCH,To High | 1 | 0 | 0 | 1
  MCV,To Low | 0 | 0 | 0 | 0
  MCV,To High | 0 | 0 | 0 | 1
  Monocytes,To Low | 2 | 3 | 1 | 0
  Monocytes,To High | 0 | 0 | 0 | 1
  Total Neutrophils,To Low | 0 | 0 | 0 | 0
  Total Neutrophils,To High | 4 | 1 | 2 | 1
  Platelet count,To Low | 1 | 0 | 1 | 0
  Platelet count,To High | 0 | 1 | 1 | 0
  RBC,To Low | 0 | 0 | 0 | 0
  RBC,To High | 0 | 1 | 0 | 1
  WBC,To Low | 1 | 0 | 0 | 0
  WBC,To High | 4 | 2 | 2 | 1

28. Secondary Outcome: Number of Participants With Worst Case Chemistry Results Post-Baseline Relative to Baseline
Description: Blood samples were collected to analyze the following Chemistry parameters: Albumin, Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Direct Bilirubin, Total Bilirubin, Calcium, C-Reactive protein, Creatinine, Glucose, Potassium, Sodium, Total Protein and Urea/Blood urea nitrogen. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose lab value category was unchanged e.g. High to High), or whose value became normal, were not recorded. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. The value at Screening was considered as Baseline. Data for Worst Case Laboratory chemistry values Post-Baseline Relative to Baseline has been presented.
Time Frame: Baseline (Screening) and up to 14 weeks
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Via DISKUS | NEMI 1000 mcg Via DISKUS | Placebo Via ELLIPTA | NEMI 700 mcg Via ELLIPTA
Number analyzed (Participants) | 14 | 14 | 8 | 8
Participants
  Albumin,To Low | 0 | 0 | 1 | 0
  Albumin,To High | 0 | 0 | 0 | 0
  ALP,To Low | 0 | 0 | 0 | 0
  ALP,To High | 0 | 0 | 0 | 1
  ALT,To Low | 0 | 0 | 0 | 0
  ALT,To High | 1 | 0 | 1 | 1
  AST,To Low | 0 | 0 | 0 | 0
  AST,To High | 0 | 0 | 0 | 0
  Direct Bilirubin,To Low | 0 | 0 | 0 | 0
  Direct Bilirubin,To High | 0 | 0 | 0 | 0
  Total Bilirubin,To Low | 0 | 0 | 0 | 0
  Total Bilirubin,To High | 1 | 0 | 0 | 0
  Calcium,To Low | 0 | 0 | 0 | 0
  Calcium,To High | 0 | 0 | 0 | 0
  C-Reactive protein,To Low | 0 | 0 | 0 | 0
  C-Reactive protein,To High | 4 | 5 | 3 | 0
  Creatinine,To Low | 1 | 0 | 1 | 0
  Creatinine,To High | 0 | 1 | 1 | 1
  Glucose,To Low | 1 | 1 | 1 | 0
  Glucose,To High | 3 | 2 | 2 | 0
  Potassium,To Low | 0 | 0 | 0 | 0
  Potassium,To High | 0 | 0 | 1 | 0
  Sodium,To Low | 0 | 2 | 2 | 0
  Sodium,To High | 0 | 0 | 0 | 0
  Total Protein,To Low | 1 | 1 | 0 | 0
  Total Protein,To High | 0 | 0 | 0 | 0
  Urea/BUN,To Low | 1 | 0 | 0 | 0
  Urea/BUN,To High | 0 | 0 | 1 | 1

29. Secondary Outcome: Number of Participants With Worst Case Vital Sign Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Vital signs were measured in semi-supine position after 5 minutes rest and included Systolic blood pressure (SBP), Diastolic blood pressure (DBP), Heart rate (HR). Data for number of participants with Post-Baseline worst case Vital Sign results relative to PCI Criteria relative to Baseline was presented. PCI ranges were: SBP (lower: <85 and upper: >160 mmHg), DBP (lower: <45 and upper: >100 mmHg), and HR (lower: <40 and upper: >110 bpm). The value at Screening was considered as Baseline.
Time Frame: Baseline (Screening) and up to 14 weeks
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Via DISKUS | NEMI 1000 mcg Via DISKUS | Placebo Via ELLIPTA | NEMI 700 mcg Via ELLIPTA
Number analyzed (Participants) | 14 | 14 | 8 | 8
Participants
  SBP, To Low | 0 | 0 | 0 | 0
  SBP, To High | 0 | 0 | 0 | 2
  DBP, To Low | 0 | 0 | 0 | 0
  DBP, To High | 0 | 0 | 0 | 0
  HR, To Low | 0 | 0 | 0 | 0
  HR, To High | 2 | 1 | 0 | 1

30. Secondary Outcome: Number of Participants With Worst Case Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: A Single 12-lead ECGs was obtained at screening and at each other timepoint during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected using the Fridericia's formula (QTcF) intervals. Data for number of participants with worst case post-Baseline abnormal ECG findings was reported. The value at Screening was considered as Baseline.
Time Frame: Up to 14 weeks
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Via DISKUS | NEMI 1000 mcg Via DISKUS | Placebo Via ELLIPTA | NEMI 700 mcg Via ELLIPTA
Number analyzed (Participants) | 14 | 14 | 8 | 8
Participants
  Abnormal - not clinically significant | 10 | 7 | 6 | 7
  Abnormal - clinically significant | 0 | 0 | 1 | 0

31. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward medical occurrence that at any dose, resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, is associated with liver injury and impaired liver function or any other situation according to medical or scientific judgment was categorized as SAE. Number of participants with AEs and SAEs have been reported.
Time Frame: Up to 14 weeks
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Via DISKUS | NEMI 1000 mcg Via DISKUS | Placebo Via ELLIPTA | NEMI 700 mcg Via ELLIPTA
Number analyzed (Participants) | 14 | 14 | 8 | 8
Participants
  Any AE | 11 | 11 | 5 | 5
  Any SAE | 2 | 3 | 4 | 0

32. Secondary Outcome: Maximum Plasma Concentration (Cmax) Following Administration of NEMI
Description: Blood samples for pharmacokinetic (PK) analysis was collected at the indicated time points following administration of NEMI via DISKUS and ELLIPTA.
Time Frame: Day 1: 5 minutes Post-dose on Day 1
Population: Pharmacokinetic Population comprised of participants in all subject population for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | NEMI 1000 mcg Via DISKUS | NEMI 700 mcg Via ELLIPTA
Number analyzed (Participants) | 14 | 7
Picograms per milliliter | 508.4 (69) | 1103.4 (34)

33. Secondary Outcome: Trough Concentration Following Administration of NEMI
Description: as for outcome 32
Time Frame: Day 1: 24 Hours post-dose; Days 12, 28, 56, 84: Pre-dose
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | NEMI 1000 mcg Via DISKUS | NEMI 700 mcg Via ELLIPTA
Number analyzed (Participants) | 14 | 8
Picograms per milliliter
  Day 1,24 hour, n=8,2: number analyzed (Participants) | 8 | 2
  Day 1,24 hour, n=8,2 | 313.9 (61) | NA (NA) — Full summary statistics are only calculated if there are 3 or more quantifiable values. There were only 2 evaluable participants in this arm for this time point and therefore data was not available.
  Day 12,pre-dose,n=9,5: number analyzed (Participants) | 9 | 5
  Day 12,pre-dose,n=9,5 | 1097.1 (38) | 1077.2 (23)
  Day 28,pre-dose, n=9,7: number analyzed (Participants) | 9 | 7
  Day 28,pre-dose, n=9,7 | 1194.3 (76) | 1225.8 (50)
  Day 56,pre-dose,n=11,7: number analyzed (Participants) | 11 | 7
  Day 56,pre-dose,n=11,7 | 1155.1 (60) | 1171.6 (49)
  Day 84,pre-dose,n=11,7: number analyzed (Participants) | 11 | 7
  Day 84,pre-dose,n=11,7 | 1339.6 (53) | 1058.2 (33)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the start of study treatment until the follow up (Up to 14 weeks)
Description: All Subjects Population was used to collect Adverse events.
Arm/Group | Placebo Via DISKUS | NEMI 1000 mcg Via DISKUS | Placebo Via ELLIPTA | NEMI 700 mcg Via ELLIPTA
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/14 | 3/14 | 4/8 | 0/8
Other Adverse Events (participants affected / at risk) | 10/14 | 10/14 | 5/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Via DISKUS (N=14) | NEMI 1000 mcg Via DISKUS (N=14) | Placebo Via ELLIPTA (N=8) | NEMI 700 mcg Via ELLIPTA (N=8)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Via DISKUS (N=14) | NEMI 1000 mcg Via DISKUS (N=14) | Placebo Via ELLIPTA (N=8) | NEMI 700 mcg Via ELLIPTA (N=8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (10) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT02522299/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT02522299/SAP_001.pdf